

#### **Protocol**

NCT Number: NCT05098041

Title: Phase 1 Open-Label Study to Evaluate the Drug-Drug Interaction of Rifampin as a Strong CYP3A Inducer on Soticlestat Pharmacokinetics in Healthy Adult

Participants

Study Number: TAK-935-1009

Document Version and Date: Final / 20 August 2021

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view with a black bar) to protect either personally identifiable information or company confidential information.

# TAKEDA PHARMACEUTICALS

Strong CYP3A Inducer on Soticlestat Pharmacokinetics in Healthy Adult Participants ne. only and Subject to the Applicable Term.

As a cipants.

Inc. only and Subject to the Applicable Term.

Percial Use only and Subject to the Applicable Term.

**Study Identifier:** TAK-935-1009

Compound: Soticlestat (TAK-935)

Takeda Development Center Americas, Inc. **Sponsor:** 

> 95 Hayden Avenue Lexington, MA 02421

Date: 20 August 2021

Final Protocol Version/Amendment

**Number:** 

# CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered. Furthermore, the information is only meant for review and compliance by the recipient, his or her brobeith of Lakega, vicabi staff, and applicable institutional review committee and regulatory agencies to enable conduct of the study.

| IAI | BLE OF CONTENTS | |
|---|---|---|
| 1.0 | STUDY SUMMARY | 6 |
| 2.0 | STUDY SCHEMATIC | |
| 3.0 | SCHEDULE OF STUDY PROCEDURES | 12 |
| 4.0 | SCHEDULE OF STUDY PROCEDURESINTRODUCTION | 15 |
| 4 | 4.1 Background | 15 |
| | INTRODUCTION. 4.1 Background 4.1.1 Soticlestat (TAK-935) | |
| | 4.1.2 Rifampin | 16 |
| 4 | 4.2 Rationale for the Proposed Study | 17 |
| 4 | 4.3 Benefit/Risk Profile | 18 |
| 5.0 | STUDY OBJECTIVES AND ENDPOINTS | 18 |
| 4 | 5.1 Hypothesis | 18 |
| | 5.2 Study Objectives | 19 |
| | 5.2.1 Study Primary Objective | 19 |
| | 5.2.2 Study Secondary Objective | 19 |
| | 5.2.3 Study Exploratory Objectives | 19 |
| - | 5.3 Endpoints | 19 |
| | 5.3.1 Primary Endpoint | 19 |
| | 5.3.2 Secondary Endpoints | 19 |
| | 5.3.3 Exploratory Endpoints | 19 |
| 6.0 | STUDY DESIGN AND DESCRIPTION | 20 |
| ( | 6.1 Study Design | |
| ( | 6.2 Dose Escalation | |
| ( | 6.3 Stopping Rules | 21 |
| ( | 6.4 Rationale for Study Design, Dose, and Endpoints | 21 |
| | 6.4.1 Rationale of Study Design. | 21 |
| | 6.4.2 Rationale for Dose | 21 |
| | 6.4.3 Rationale for Endpoints | 21 |
| | 6.4.4 Future Biomedical Research | 22 |
| (KK | 6.4.5 Critical Procedures Based on Study Objectives: Timing of Proced | lures22 |
| 3) | 6.5 Study Design/Dosing/Procedures Modifications Permitted Within Pro | |
| | Parameters | |
| ( | 6.6 Study Beginning and End/Completion | |
| | 6.6.1 Definition of Beginning of the Study | 22 |
| | 6.6.2 Definition of End of the Study | 22 |

| | 6.6.3 | Definition of Study Completion | .22 |
|---|---|---|---|
| | 6.6.4 | Definition of Study Discontinuation | .23 |
| | 6.6.5 | Criteria for Premature Termination or Suspension of the Study | |
| | 6.6.6 | | .23 |
| 7.0 | SELEC | CTION AND DISCONTINUATION/WITHDRAWAL OF PARTICIPANTS | .23 |
| 7.1 | Inc | Plusion Criteria | .23 |
| 7.2 | 2 Ex | clusion Criteria | .24 |
| 7.3 | B Ex | clusion Criteria cluded Medications, Supplements, Dietary Products et, Fluid, Activity Diet and Fluid | .25 |
| 7.4 | l Di | et, Fluid, Activity | .27 |
| | 7.4.1 | Diet and Fluid | .27 |
| | 7.1.2 | | . 20 |
| 7.5 | 5 Cr | iteria for Discontinuation or Withdrawal of a Participant | .28 |
| 7.6 | 5 Pro | ocedures for Discontinuation or Withdrawal of a Participant | .29 |
| 7.7 | | rticipant Replacement | |
| 8.0 | CLINI | CAL STUDY MATERIAL MANAGEMENT | .30 |
| 8.1 | Cli | inical Study Drug | .30 |
| | 8.1.1 | Clinical Study Drug Labeling | .30 |
| | 8.1.2 | Clinical Study Drug Inventory and Storage | .30 |
| | 8.1.3 | Clinical Study Drug Blinding | .30 |
| | 8.1.4 | Randomization Code Creation and Storage | .31 |
| | 8.1.5 | Clinical Study Blind Maintenance/Unblinding Procedure | .31 |
| | 8.1.6 | Accountability and Destruction of Sponsor-Supplied Drugs | .31 |
| 9.0 | STUD | Y PROCEDURES | .31 |
| 9.1 | Ad | Iministrative Procedures | .31 |
| | 9.1.1 | Informed Consent Procedure | .31 |
| | 9.1.2 | Inclusion and Exclusion | .31 |
| | 9.1.3 | Medical History/Demography | .32 |
| | 9.1.4 | Concomitant Medications | .32 |
| 9.2 | Cli | inical Procedures and Assessments | .32 |
| ,01 | 9.2.1 | Physical Exam | .32 |
| Sign | 9.2.2 | Height and Weight | .32 |
| | 9.2.3 | BMI | .32 |
| | 9.2.4 | Vital Signs | .33 |
| | 9.2.5 | 12-Lead ECG | .33 |
| | 9.2.6 | Study Drug Administration | .33 |

| 9.2.7 C-SSRS | 34 |
|---|---|
| 9.2.8 AE Monitoring | 34 |
| 9.2.9 Laboratory Procedures and Assessments | 34 |
| 9.3 Pharmacokinetic Samples | 88 <sub>2221</sub> |
| 0.0.4 701 11 11 11 11 11 | |
| 9.3.2 Biomarker Measurements | 37 |
| 9.3.3 PGx Measurements | 38 |
| 9.3.1 Pharmacokinetic Measurements 9.3.2 Biomarker Measurements 9.3.3 PGx Measurements 9.3.4 Confinement 10.0 ADVERSE EVENTS 10.1 Definitions and Elements of AEs 10.1.1 SAEs 10.1.2 Special Interest AEs 10.2 AE Procedures 10.2.1 Assigning Severity/Intensity of AEs 10.2.2 Assigning Causality of AEs 10.2.3 Start Date 10.2.4 End Date | 38 |
| 10.0 ADVERSE EVENTS | |
| 10.1 Definitions and Elements of AEs | |
| 10.1.1 SAEs | 40 |
| 10.1.2 Special Interest AEs | 41 |
| 10.2 AE Procedures | 41 |
| 10.2.1 Assigning Severity/Intensity of AEs | 41 |
| 10.2.2 Assigning Causality of AEs | 42 |
| 10.2.3 Start Date | 42 |
| 10.2.4 End Date | 42 |
| 10.2.5 Tattern of Maverse Event (Trequency) | |
| 10.2.6 Action Taken With Study Treatment | 43 |
| 10.2.7 Outcome | 43 |
| 10.2.8 Collection and Reporting of AEs, SAEs, Special | Interest AEs, and Abnormal |
| LFTs | 43 |
| 10.2.9 Safety Reporting to Investigators, IRBs or IECs | |
| 11.0 STATISTICAL METHODS | |
| 11.1 Statistical and Analytical Plans | |
| 11.1.1 Apalysis Sets | |
| 11.1.2 Analysis of Demography and Other Baseline Ch | |
| 11.03 PK Analysis | |
| 19.1.4 PD Analysis | |
| 11.1.5 Safety Analysis | |
| 11.2 Interim Analysis and Criteria for Early Termination | |
| 11.3 Determination of Sample Size | |
| 12.0 QUALITY CONTROL AND QUALITY ASSURANCE | |
| 12.1 Study-Site Monitoring Visits | |
| 12.2 Protocol Deviations | |
| 12.3 Quality Assurance Audits and Regulatory Agency In | nspections49 |

| 13.0 ETHIC | CAL ASPECTS OF THE STUDY | 50 |
|---|---|---|
| 13.1 IR | B and/or IEC Approval | 50 |
| 13.2 Par | rticipant Information, Informed Consent, and Participant Authorization | 51 |
| 13.3 Par | rticipant Confidentiality | 52 |
| 13.4 Pu | rticipant Confidentialityblication, Disclosure, and Clinical Study Registration Policy | 52 |
| 13.4.1 | Publication and Disclosure | 52 |
| 13.4.2 | Clinical Study Registration. | 53 |
| 13.4.3 | Clinical Study Results Disclosure | 53 |
| 13.5 Ins | surance and Compensation for Injury | 53 |
| 14.0 ADMI | Publication and Disclosure Publication and Disclosure Clinical Study Registration Clinical Study Results Disclosure Surance and Compensation for Injury NISTRATIVE AND REFERENCE INFORMATION Iministrative Information Study Contact Information INVESTIGATOR AGREEMENT Study-Related Responsibilities List of Abbreviations HANDLING AND RECORD KEEPING RFs (Electronic and Paper) Cord Retention | 53 |
| 14.1 Ad | ministrative Information | 53 |
| 14.1.1 | Study Contact Information | 54 |
| 14.1.2 | INVESTIGATOR AGREEMENT | 55 |
| 14.1.3 | Study-Related Responsibilities | 56 |
| 14.1.4 | List of Abbreviations | 56 |
| 15.0 DATA | HANDLING AND RECORD KEEPING | 57 |
| 15.1 CR | RFs (Electronic and Paper) | 57 |
| 15.2 Re | cord Retention | 58 |
| 16.0 REFEI | RENCES | 59 |
| 17.0 APPE | NDICES | 60 |
| | cord Retention RENCES NDICES | |
| I IST OF IN | TEXT TABLES | |
| | | 11 |
| Table 2.a | Study Schematic Dose Regimens for Study Drugs | |
| Table 2.b Table 7.a | | |
| | Excluded Medications, Supplements, and Dietary Products | |
| | Primary Specimen Collections | |
| Table 10.a | Takeda Medicany Significant AE List | 41 |
| LIST OF AP | PENDICES | |
| Appendix A | Responsibilities of the Investigator | 60 |
| Appendix B | Elements of the Participant Informed Consent | |
| Appendix C | Investigator Consent to the Use of Personal Information | |
| Appendix D | Pregnancy and Contraception | 66 |

#### 1.0 STUDY SUMMARY

| Name of Sponsor: | Compound: |
|-------------------------------------------------|-----------------------|
| Takeda Development Center Americas, Inc. (TDCA) | Soticlestat (TAK-935) |
| 95 Hayden Avenue | |
| Lexington, MA 02421 | 70' |
| Telephone: +1 (617) 679-7000 | <b>%</b> 0 |
| Study Identifier: TAK-935-1009 | Phase: 1 |

**Protocol Title:** A Phase 1 Open-Label Study to Evaluate the Drug-Drug Interaction of Rifampin as a Strong CYP3A Inducer on Soticlestat Pharmacokinetics in Healthy Adult Participants

#### **Study Design:**

This is an open-label, 2-period, fixed-sequence drug-drug interaction (DDI) study to evaluate the effect of a strong cytochrome P450 (CYP) 3A inducer, rifampin, on the single-dose pharmacokinetics (PK) of soticlestat in healthy participants.

Study schematic of the study design and dose regimens are shown in Table 2a and Table 2.b. A schedule of assessments is shown in Schedule of Study Procedures (Section 3.0).

Participants will be screened within 4 weeks (28 days) prior to the first administration of soticlestat (Day -28 to first dosing, Day 1). Qualified participants will be admitted to the clinic on Day -1 of Period 1, at the time indicated by the Clinical Research Unit (CRU), and will remain confined until after the last blood draw and/or study procedures on Day 14 of Period 2.

In Period 1, on Day 1, participants will receive a single **oral** dose of soticlestat (300 mg; 3 x 100 mg immediate-release tablets [T4 tablets]) under fasting conditions. **Blood** samples for the PK of soticlestat will be collected at scheduled time points from predose through 96 hours postdose. There will be washout period of 4 days between the soticlestat dose in Period 1 and the first rifampin dose in Period 2.

In Period 2, from Days 1 to 13, participants will receive a once daily (QD) oral dose of rifampin (600 mg; 2 x300 mg capsules) under fasting conditions. On the morning of Day 11, participants will receive a single dose of soticlestat (300 mg; 3 x 100 mg T4 tablets) co-administered with the rifampin dose under fasting conditions. Blood samples for the PK of soticlestat will be collected at scheduled time points from soticlestat predose on Day 11 through 72 hours postdose.

Safety and tolerability will be assessed throughout the study by treatment-emergent adverse events (TEAEs), clinical laboratory evaluations, physical examinations, 12-lead electrocardiograms (ECGs), vital signs, and Columbia-Suicide Severity Rating Scale (C-SSRS).

After discharge, the CRU will contact all participants (including participants who terminate the study early) 15 ( $\pm$  2) days after the last soticlestat administration by telephone or other methods per CRU standards to determine if any adverse event (AE) has occurred or concomitant medications have been taken since the last study visit. If clinically significant findings are observed upon discharge, participants may return to the CRU for re-evaluation per Investigator's discretion.

#### **Study Primary Objective:**

To characterize the effect of rifampin, a strong CYP3A inducer, on the single-dose PK of soticlestat.

#### **Study Secondary Objective:**

To assess the safety and tolerability of soticlestat following a single oral dose in healthy adult participants with/without a strong CYP3A inducer.

| Study Participants Population: Healthy male and female participal | pants aged 18 to 55 years inclusive, at screening. |
|---|---|
| Body Mass Index (BMI) 18.0-32.0 kg/m <sup>2</sup> , inclusive, at screening | ico |

| Dody Mass mack (DMH) 10.0-32.0 kg/m, metasive, at | screening |
|---|---|
| Planned Number of Participants: | Planned Number of Sites: |
| 14 participants will be enrolled | 1 |
| Dose Levels: | Route of Administration: |
| Soticlestat | Oral |
| 300 mg (3 x 100 mg strength T4 tablets) | C. |
| Rifampin | 30 |
| 600 mg (2 x 300 mg strength capsules) | Sur |
| Duration of Treatment: | Planned Study Duration: |
| Soticlestat: Single dose on Day 1 Period 1 and on Day | Approximately 58 days including screening and follow-up. |
| 11 Period 2. | 41 |
| Rifampin: QD for 13 consecutive days (Days 1-13) | O, |
| Period 2. | |

#### **Criteria for Inclusion:**

Participants must fulfill the following inclusion criteria before the first dose to be eligible for participation in the study:

- 1. Healthy, adult, male or female of non-childbearing potential (Appendix D), 18 55 years of age, inclusive, at screening.
- 2. Male participant agrees to comply with any applicable contraceptive requirements of the protocol as detailed in Appendix D.
- 3. BMI  $\ge$ 18.0 and  $\le$ 32.0 kg/m<sup>2</sup> at screening.
- 4. Continuous non-smoker who has not used nicotine-containing products for at least 90 days prior to the first dosing.
- 5. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs, as deemed by the PI or designee.
  - Supine BP is ≥90/40 mmHg and ≤140/90 mmHg at screening;
  - Supine PR is  $\ge$ 45 bpm and  $\le$ 100 bpm at screening;
  - QTcF is  $\leq$ 450 msec (males) or  $\leq$ 470 msec (females) and ECG findings considered normal or not clinically significant by the Investigator or designee at screening;
  - Estimated creatinine clearance ≥80 mL/min at screening;
  - Liver function tests including alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 X the upper limit of normal (ULN) at screening and check-in.
- 6. Able to swallow multiple tablets/capsules.
- 7. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

#### **Criteria for Exclusion:**

Participants must not be enrolled in the study if they meet any of the following criteria before the first dose of study drug:

- 1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
- 2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
- 3. History or presence of gastritis, gastrointestinal tract, gastric bypass surgery, or hepatic disorder or other clinical condition which, in the opinion of the Investigator or designee, may affect the absorption, distribution, metabolism, or elimination of study drugs.
- 4. History or presence of cataracts or other clinically significant vision disturbances.
- 5. History or presence of epilepsy, seizure, or convulsion, tremor or related symptoms.
- 6. History of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
- 7. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
- 8. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
- 9. Any positive responses on the C-SSRS that in the clinical judgment of the Investigator has a risk of suicide or has made a suicide attempt in the previous 12 months prior to the first dosing.
- 10. Female participants of childbearing potential.
- 11. Female participants with a positive pregnancy test at screening or check-in or who is lactating.
- 12. Positive urine drug or alcohol results at screening or check-in.
- 13. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
- 14. Unable to refrain from or anticipates the use of:
  - Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to first dosing.
- 15. History of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to the following: beer [354 mL/12 oz], wine [118 mL/4 oz], or distilled spirits [29.5 mL/1 oz] per day).
- 16. Consumes excessive amounts, defined as greater than 4 servings (1 serving is approximately equivalent to 120 mg of caffeine), of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
- 17. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
- 18. Donation of blood or significant blood loss within 56 days prior to the first dosing.
- 19. Plasma donation within 7 days prior to the first dosing.
- 20. Participation in another clinical study within 30 days or 5 half-lives prior to the first dosing. The 30-days window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

# Main Criteria for Evaluation and Analyses:

Primary Endpoints:

The following PK parameters will be analyzed for soticlestat, when administered alone and when co-administered with rifampin:

- Maximum observed concentration ( $C_{max}$ ).
- Area under the concentration-time curve from time 0 to infinity, calculated using the observed value of the

last quantifiable concentration (AUC $_{\infty}$ ).

- Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration
- Time of first occurrence of  $C_{max}$  ( $t_{max}$ ).

#### Secondary Endpoint:

- Number of participants with at least one TEAE.
- Incidence of clinically significant abnormal values for laboratory evaluations, vital signs, ECG parameters, and C-SSPS and C-SSRS.

## **Statistical Considerations:**

Pharmacokinetics:

Natural log (ln)-transformed AUC<sub>last</sub>, AUC<sub>o</sub>, and C<sub>max</sub> data will be analyzed using a linear mixed effects model, separately. The model will include treatment (soticlestat with and without rifampin) as a fixed effect and participant as a random effect. The point estimate and 90% confidence interval (CI) for the geometric mean ratio (GMR) of AUC<sub>∞</sub> for the soticlestat with versus without rifampin will be calculated. The same approach will be used to estimate the GMR of AUC<sub>last</sub> and C<sub>max</sub> of soticlestat with versus without rifampin.

The same analysis as described above will be conducted for soticlestat metabolites if appropriate.

Safety:

AEs will be tabulated. Summary statistics for vital signs, safety 12-lead ECGs, C-SSRS, and clinical laboratory Property of Taked assessments will be computed and provided.

## **Sample Size Justification:**

This study is not powered for hypothesis testing and is not based on any specific no-effect boundaries. The sample size is based on an estimation approach and is considered sufficient to provide a reliable estimate of the DDI magnitude.

s. comple subject to the state of the state A total of 14 participants will be dosed to ensure that 12 evaluable subjects complete the study.

#### 2.0 STUDY SCHEMATIC

Table 2.a **Study Schematic** 

| | | Period 1 | | | 1 SILL | | |
|---|---|---|---|---|---|---|---|
| Screening | Check-in and<br>Predose<br>Assessments | Soticlestat<br>Dosing, PK<br>Sampling,<br>and Study<br>Assessments | PK Sampling<br>and Study<br>Assessments | Rifampin<br>Dosing and<br>Study<br>Assessments | Co-administration<br>(Rifampin and<br>Soticlestat), PK<br>Sampling, and<br>Study Assessments | Rifampin<br>Dosing, PK<br>Sampling and<br>Study<br>Assessments | |
| Within<br>28 days<br>prior to first<br>dosing | Day -1 | Day 1 | Day 2-5 <sup>a</sup> | Day 1ª-10 | Day 11 110 | Day 12 -14 <sup>c</sup> | 15 (± 2)<br>days<br>following<br>last<br>soticlestat<br>dose |
| | | | Confine | ment <sup>b</sup> | | | Contact |

| | Study Drug | Dose | Dose Regimen | Number of Days on Study Drug |
|---|---|---|---|---|
| | Soticlestat (T4 tablets) | 300 mg<br>(3 x 100 mg<br>tablets) | Single dose, oral | Day 1 Period 1 and Day 11 Period 2 |
| | Rifampin (capsules) | 600 mg<br>(2 x 300 mg<br>capsules) | QD, oral | Days 1 through 13 Period 2 |
| Prof | perty of Lakeda. Fo | , Non' | | |

Day 5 Period 1 will also be considered Day 1 Period 2.

b Participants will start the confinement on Day -1 Period 1 and will remain confined until Day 14 Period 2.

c Last dose of rifampin will be administered on Day 13.

Table 2.b Dose Regimens for Study Drugs

# 3.0 SCHEDULE OF STUDY PROCEDURES

| Study Procedures <sup>a</sup> | | | Study Days in Period 1 ° | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days in Period → | S b | -1 | | | | | | | 1 | | | | 20 | 7 | | 2 | , | 3 | 4 | 5 |
| Hours → | | C-I d | 0 | 0.133 | 0.25 | 0.5 | 0.75 | 1 | 1.5 | 2 | 4 | 6 | 8 | 10 | 14 | 24 | 36 | 48 | 72 | 96 e |
| Administrative Procedures | | | | | | | | | | | | 110 | , | | | | | | | |
| Informed Consent | X | | | | | | | | | | × | 0 | | | | | | | | |
| Inclusion/Exclusion Criteria | X | X | | | | | | | | | -C) | | | | | | | | | |
| Medical History | X | | | | | | | | | Ś | 0 | | | | | | | | | |
| Safety Evaluations | | | | | | | | | | 301 | | | | | | | | | | |
| Physical Examination <sup>f</sup> | X | X | | | | | | | 7 | | | | | | | | | | | |
| Height | X | | | | | | | | | | | | | | | | | | | |
| Weight | X | | | | | | | 14 | 0 | | | | | | | | | | | |
| 12-Lead Safety ECG <sup>g</sup> | X | X¹ | | | | | | 16, | | | | | | | | | | | | |
| Vital Signs (PR, BP, RR, and T) g | X | X¹ | | | | X | -01 | | X | | | | | | | X | | | | |
| Hem, Coag, Serum Chem h, and UA | X | X | | | | , | 3 | | | | | | | | | | | X | | |
| Serum Pregnancy Test (♀ only) | X | X | | | | | | | | | | | | | | | | | | |
| Serum FSH (♀ only) | X | | | | ٠, ( | 30 | | | | | | | | | | | | | | |
| Urine Drug and Alcohol Screen | X | X | | | VO. | | | | | | | | | | | | | | | |
| HIV/Hepatitis B and C Screen | X | | | 2 | | | | | | | | | | | | | | | | |
| C-SSRS J | X | X | | C'O, | | | | | | | | | | | | | | | | |
| AE Monitoring | | | · C | 7 | | | | | | Σ | ζ | | | | | | | ı | | |
| ConMeds Monitoring | | X | | | | | | | | | | | | | | | | | | |
| Study Drug Administration / PK | | Z) | | | | | | | | | | | | | | | | | | |
| Soticlestat Administration | | ₹\bar{\bar{\bar{\bar{\bar{\bar{\bar{ | X k | | | | | | | | | | | | | | | | | |
| Blood for Soticlestat | 9 | <b>)</b> | X 1 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X 1 |
| Other Procedures | | | | | | | | | | | | | | | | | | | | |
| Confinement in the CRU <sup>d</sup> | | | | | | | | | | | X | | | | | | | | | |

Page 13 of 67 20 August 2021

| Study Procedures <sup>a</sup> | | Study Days in Period 2 ° | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days in Period→ | 1 e | 2 - 9 | 10 | | | 11 12 13 14 | | | | | | | | 14 | ET m | FU <sup>n</sup> | | | | | | |
| Hours → | 0 | 0 | 0 | 0 | 0.133 | 0.25 | 0.5 | 0.75 | 1 | 1.5 | 2 | 4 | 6 | 8 | 10 | 14 | 24 | 36 | 48 | 72 | | |
| Safety Evaluations | | | | | | | | | | | | | | | 2 | )4 | | | | | | |
| 12-Lead Safety ECG <sup>g</sup> | | | | X º | | | | | | | | | | _ ( | 2) ( | | | | | X | X | |
| Vital Signs (PR, BP. RR, and T) <sup>g</sup> | | | | Xº | | | X | | | X | | | | 11. | | | $X^{1}$ | | | X | X | |
| Hem, Serum Chem <sup>h</sup> , and UA | | | | Xº | | | | | | | | | , × | O | | | | | $X^{\perp}$ | | X | |
| C-SSRS J | | | | | | | | | | | | | CO. | | | | | | | X | X | |
| AE Monitoring | | | X | | | | | | | | | | | | | | | | | | | |
| ConMeds Monitoring | | | | | | | | | | | 2 | 50, | | | | | | | | | | X |
| Study Drug Administration / PK | | | | | | | | | | | Dilli | | | | | | | | | | | |
| Rifampin Administration p | X | X | X | X | | | | | | 17 | J | | | | | | X | | X | | | |
| Soticlestat Administration | | | | X k | | | | | | 6, | | | | | | | | | | | | |
| Blood for Soticlestat | | | | X 1 | X | X | X | X | °x | X | X | X | X | X | X | X | X 1 | X | X 1 | X | X | |
| Other Procedures | | | | | | | | 9, | | | | | | | | | | | | | | |
| Confinement in the CRU d | | • | | | | | NO. | | | X | | • | | • | • | • | | • | | | | |

- a. For details on Procedures, refer to Section 9.0.
- b. Within 28 days prior to the first dosing.
- c. There will be washout period of 4 days between the soticlestat dose in Period 1 and the first rifampin dose in Period 2.
- d. Participants will be admitted to the CRU on Day -1 of Period 1, at the time indicated by the CRU, and be confined throughout the study (Day 14 of Period 2). Participants may be asked to check-in to the CRU earlier to undergo additional COVID-19 precaution procedures.
- e. Day 5 of Period 1 will be the same as Day 1 of Period 2, study procedures scheduled for both days will only be performed once.
- f. A full physical examination will be conducted at screening. An abbreviated physical examination will be conducted at check-in. Symptom-driven physical examinations may be performed during the study, at the Investigator's or designee's discretion.
- g. All assessments will be performed after participants have rested for at least 5 minutes in the supine position.
- h. Samples for serum chemistry will be obtained following a fast of at least 8 hours, however, in case of dropouts or rechecks, participants may not have fasted for 8 hours prior to when the serum chemistry sample is taken.
- i. To be performed within 24 hours prior to dosing of soticlestat.

CONFIDENTIAL

- j. At screening, the C-SSRS Baseline/Screening version will be administered; at all other time points, the Since Last Visit version will be administered.
- k. Soticlestat will be administered after an overnight fast of at least 10 hours. Fasting will continue for at least 4 hours postdose.
- 1. To be performed prior to dosing.
- m. To be performed prior to early termination from the study.
- n. The CRU will contact all participants (including participants who terminate the study early) 15 ( $\pm$  2) days after the last soticlestat administration by telephone or other methods per CRU standards to determine if any AE has occurred since the last study visit.
- o. To be performed within 2 hours prior to dosing of soticlestat.
- p. On Day 11 (Period 2), participants will receive soticlestat and rifampin together, after an overnight fast of at least 10 hours. On Days 1 to 10 and Days 12 and 13 (Period2), rifampin will be administered after an overnight fast of at least 8 hours. No food is allowed during the first 4 hours after drug administration.

Abbreviations: ♀ = Females, AE = Adverse events, BP = Blood pressure, C-I = Check-in, C-SSRS = Colombia-Suicide Severity Rating Scale Chem = Chemistry, Coag = Coagulation, ConMeds = Concomitant medication, CRU = Clinical research unit, ECG = Electrocardiogram, ET = Early termination, FSH = Follicle-stimulating hormone, FU = Follow-up, Hem = Hematology, HIV = Human immunodeficiency virus, PK = Pharmacokinetics, PR = Pulse rate, RR = Respiratory rate, S = Screening, T = Temperature, UA = Urinalysis.

#### 4.0 INTRODUCTION

#### 4.1 **Background**

#### **Soticlestat (TAK-935)** 4.1.1

ims of Use Soticlestat is a potent and selective cholesterol 24S hydroxylase (CH24H) inhibitor currently in development as an oral adjunct to standard of care therapy for the treatment of rare pediatric epilepsies referred to as Developmental and Epileptic Encephalopathies (DEE) which is a cluster of pediatric epilepsy syndromes and includes Dravet Syndrome (DS) and Lennox Gastaut Syndrome (LGS). Epilepsy is linked to a dysregulation in glutamatergic signaling brought upon by an over-activation of CH24H. This enzyme is predominantly expressed in neurons and involved in the homeostasis of brain cholesterol by converting it to 245-hydroxycholesterol, a polar metabolite capable of passing the blood-brain barrier via lipoproteins.

Soticlestat is a first-in-class therapeutic candidate that has the potential to control seizures in treatment-resistant patients with epilepsy by reducing over-activated glutamate signaling modulating reactive astrocytes and reducing over-activated glutamate signaling in neurons. This mechanism of action is thought to clinically manage seizures by reducing seizure frequency and severity as well as brain damage and cognitive deficits that are pathological sequelae of the epileptogenic process but also other conditions where excessive glutamatergic signaling activity drives the pathology.



# **Clinical Safety and Pharmacokinetics**

The PK, safety, tolerability, and efficacy of soticlestat have been evaluated in 6 phase 1 clinical studies in healthy participants (completed), a phase 1b/2a in participants with DEEs (completed), and 2 phase 2 studies in participants with DS, LGS, 15q11-q13 duplication syndrome (Dup15q), or CDKL5 deficiency disorder (CDD; clinically completed [study completed, clinical study report (CSR) pending]). One phase 2, open-label, long-term study in participants with various

DEEs, including DS, LGS, Dup15q, or CDD, is ongoing. In addition, 2 phase 1 studies in healthy participants and 1 phase 2 study in participants with complex regional pain syndrome (CRPS) are clinically completed with data analysis or CSR pending. Overall, 350 participants have been enrolled in the clinical trials with soticlestat, of which 310 have received active treatment based on actual exposure data from completed clinical trials and enrollment at the time of data lock point for ongoing clinical trials.

Soticlestat was rapidly absorbed with an average median  $t_{max}$  of 0.25 to 0.52 hours following single-dose (15 to 1350 mg) and an average median  $t_{max}$  of 0.33 to 0.5 hours following multiple-dose (100 to 600 mg) under fasting conditions in healthy participants. When administered under fed conditions, soticlestat  $t_{max}$  was delayed by about 1.5 hours,  $C_{max}$  was decreased by 60%, however food had little impact on the total exposure of the drug as AUC decreased by only 11% using the tablet formulation. Soticlestat was shown to cross the blood brain barrier and was able to block tracer binding to the enzyme target, demonstrating a sigmoidal maximum observed effect.

Refer to the Investigator's Brochure (IB) for detailed background information on soticlestat [2].

## 4.1.2 Rifampin

Rifampin is a semisynthetic antibiotic derivative of rifamycin SV. Rifampin inhibits deoxyribonucleic acid-dependent ribonucleic acid polymerase activity in susceptible *Mycobacterium tuberculosis* organisms [3].

After oral administration, rifampin is readily and completely absorbed from the gastrointestinal tract. Serum  $C_{max}$  in healthy adults and pediatric populations vary widely from individual to individual. After a single 600 mg oral dose of rifampin in healthy adults,  $C_{max}$  is reached within 1 - 2 hours and peak serum concentration averages at 7  $\mu$ g/mL but may vary from 4 - 32  $\mu$ g/mL. Absorption of rifampin is reduced by about 30% when the drug is ingested with food. Thus, daily doses of rifampin should be given at least 1 hour before or 2 hours after a meal [3].

After absorption, rifampin is rapidly eliminated in the bile, and an enterohepatic circulation ensues. During this process, rifampin undergoes progressive deacetylation to form the desacetylrifampin metabolite, and nearly all the drug in the bile is in this form by ~6 hours. Following multiple dosing, rifampin is a potent inducer of drug metabolism by inducing a variety of hepatic and intestinal CYP enzymes, especially CYP3A4 [3].

Systemic hypersensitivity reactions were reported with rifampin administration. Signs and symptoms of hypersensitivity reactions may include fever, rash, urticaria, angioedema, hypotension, acute bronchospasm, conjunctivitis, thrombocytopenia, neutropenia, elevated liver transaminases or flu-like syndrome (weakness, fatigue, muscle pain, nausea, vomiting, headache, chills, aches, itching, sweats, dizziness, shortness of breath, chest pain, cough, syncope, palpitations). Isolated reports have associated porphyria exacerbation with rifampin administration [3].

# 4.2 Rationale for the Proposed Study

Although metabolism via CYP3A4 is not the main route of elimination for soticlestat, there is still a potential of decrease in soticlestat systemic exposure when it is concomitantly administered with strong CYP3A inducers because of the induction of CYP3A-mediated intestinal and/or hepatic metabolism following oral dose administration of these inducers.

The purpose of this study is therefore to assess the effect of co-administration of a strong CYP3A inducer on the PK soticlestat to provide information for management of potential DDIs with strong CYP3A inducers in future clinical studies of soticlestat.

Rifampin was chosen as a perpetrator for this study as it is considered a strong index inducer of CYP3A as per the Food and Drug Administration [4]. In addition, rifampin also induces UGT1A9 and UGT2B4 [5-7] and direct glucuronidation by UGT1A9 and 2B4 is the

predominant clearance pathway of soticlestat, this study will also inform strategies for management of potential DDIs with UGT1A9 and UGT2B4 inducers in future clinical studies of soticlestat.

#### 4.3 Benefit/Risk Profile

The dose of 300 mg soticlestat is the recommended phase 3 dose [2] and will be administered as a single-dose in this study. In addition, doses up to 1350 mg were administered in healthy participants and were found to be safe and well tolerated.

The doses of rifampin are administered for a very short duration in this study, any potential risk(s) to participants in this study following cumulative intake will be mitigated according to the dosing recommendations presented in the labelling [3].



The inclusion and exclusion criteria, screening, and safety monitoring practices employed by this protocol (ie, 12-lead ECG, vital signs, clinical laboratory tests, AE questioning, C-SSRS, and physical examinations) are adequate to protect the participant's safety and should detect all TEAEs.

There will be no direct health benefit for study participants from receipt of study drugs. An indirect health benefit to the healthy participants enrolled in this study is the free medical tests received at screening and during the study.

## 5.0 STUDY OBJECTIVES AND ENDPOINTS

## 5.1 Hypothesis

Not applicable.

# 5.2 Study Objectives

# 5.2.1 Study Primary Objective

To characterize the effect of rifampin, a strong CYP3A inducer, on the single-dose PK of soticlestat.

# 5.2.2 Study Secondary Objective

To assess the safety and tolerability of soticlestat following a single oral dose in healthy adult participants with/without a strong CYP3A inducer.

# 5.3 Endpoints

## **5.3.1** Primary Endpoint

The following PK parameters will be analyzed for soticlestat, when administered alone and when co-administered with rifampin:

- Maximum observed concentration (C<sub>max</sub>).
- Area under the concentration-time curve from time 0 to infinity, calculated using the observed value of the last quantifiable concentration ( $AUC_{\infty}$ ).
- Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC<sub>last</sub>).
- Time of first occurrence of Cmax (t<sub>max</sub>).

# 5.3.2 Secondary Endpoints

- Number of participants with at least one TEAE.
- Incidence of clinically significant abnormal values for laboratory evaluations, vital signs, ECG parameters, and C-SSRS.



#### 6.0 STUDY DESIGN AND DESCRIPTION

## 6.1 Study Design

This is an open-label, 2-period, fixed sequence DDI study to evaluate the effect of a strong CYP3A inducer, rifampin, on the single-dose PK of soticlestat in healthy participants.

Study schematic of the study design and dose regimens are shown in Table 2.a and Table 2.b. A schedule of assessments is shown in Schedule of Study Procedures (Section 3.0).

Participants will be screened within 4 weeks (28 days) prior to the first administration of soticlestat (Day -28 to first dosing, Day 1). Qualified participants will be admitted to the clinic on Day -1 of Period 1, at the time indicated by the CRU, and will remain confined until after the last blood draw and/or study procedures on Day 14 of Period 2.

In Period 1, on Day 1, participants will receive a single dose of soticlestat (300 mg; 3 x 100 mg T4 tablets) under fasting conditions. Blood samples for the PK of soticlestat will be collected at scheduled time points from predose through 96 hours postdose. There will be washout period of 4 days between the soticlestat dose in Period 1 and the first rifampin dose in Period 2.

In Period 2, from Days I to 13, participants will receive a QD oral dose of rifampin (600 mg; 2 x 300 mg capsules) under fasting conditions. On the morning of Day 11, participants will receive a single dose of soticlestat (300 mg; 3 x 100 mg T4 tablets) co-administered with the rifampin dose under fasting conditions. Blood samples for the PK of soticlestat will be collected at scheduled time points from soticlestat predose on Day 11 through 72 hours postdose.

Safety and tolerability will be assessed throughout the study by TEAEs, clinical laboratory evaluations, physical examinations, 12-lead ECGs, vital signs, and C-SSRS.

After discharge, the CRU will contact all participants (including participants who terminate the study early) 15 ( $\pm$  2) days after the last soticlestat administration by telephone or other methods per CRU standards to determine if any AE has occurred or concomitant medications have been taken since the last study visit. If clinically significant findings are observed upon discharge, participants may return to the CRU for re-evaluation per Investigator's discretion.

#### 6.2 Dose Escalation

Not applicable.

## 6.3 Stopping Rules

Not applicable.

## 6.4 Rationale for Study Design, Dose, and Endpoints

# 6.4.1 Rationale of Study Design

This study will evaluate the effect of rifampin on soticlestat using an open-label, 2-period, fixed sequence. A fixed-sequence design has been selected as this will reduce the study duration and prevent any carryover effects of the study treatment. Since the absorption of rifampin is reduced when it is administered with food [3], it was thus decided to administer all study drugs under fasting conditions. The washout period of 4 days between the soticlestat dosing alone (Day 1 of Period 1) and the first rifampin dose (Day 1 of Period 2) is considered sufficient to prevent carryover effect of the treatment.

#### 6.4.2 Rationale for Dose

The dose of soticlestat selected for this study is 300 mg (3 x 100 mg), the recommended phase 3 dose. In clinical studies, soticlestat was safe and well tolerated when administered as a single dose up to 1350 mg.

The dose of rifampin selected for this study is 600 mg (2 x 300 mg) QD, which is commonly used in therapeutic regimens. The  $t_{22}$  of rifampin is ~3 hours following a 600 mg oral dose [3]; however, the time required to produce maximum enzyme induction is substantially longer due to the need for enzyme production. The timeframe for maximum induction by rifampin has been estimated as at least 5 days following administration of 600 mg QD [9-10]. In most in vivo interaction studies in healthy adult participants, oral rifampin has typically been administered as a 600 mg dose for 4 to 18 days [11]. To maximize induction of CYP3A4, rifampin will be administered QD for 10 days prior to co-administration with soticlestat on Day 11 (Period 2). To maintain the level of induction, rifampin will be administered throughout PK sampling of soticlestat (ie, until Day 13 of Period 2).

# 6.4.3 Rationale for Endpoints

# 6.4.3.1 Pharmacokinetic Endpoints

The PK endpoints are standard for this type of study.

## 6.4.3.2 Safety Endpoints

The key safety endpoints are typical for phase 1 studies and will be assessed through monitoring of AEs, vital signs, ECGs, clinical laboratory assessments, C-SSRS, and physical examinations.



# 6.4.5 Critical Procedures Based on Study Objectives: Timing of Procedures

For this study, the critical component is the blood collection for plasma concentrations of soticlestat and is to be collected as close to the scheduled times defined in this protocol as possible.

# 6.5 Study Design/Dosing/Procedures Modifications Permitted Within Protocol Parameters

The dose and administration of the study drugs to any participant may not be modified. Unscheduled procedures might be performed for safety reasons. If necessary, a participant may be discontinued for the reasons described in Section 7.5 and Section 7.6.

## 6.6 Study Beginning and End/Completion

# 6.6.1 Definition of Beginning of the Study

The beginning of the study will be defined as the beginning of the screening (ie, signing of the ICF) of the first participant.

# **6.6.2 Definition of End of the Study**

The end of study is defined as the date of the last scheduled study procedure as outlined in the Schedule of Study Procedures (Section 3.0)

## **6.6.3** Definition of Study Completion

Study completion is defined as the date when the last follow-up visit for the last participating participant in the study is completed.

ins of Use This time period may change in the event that the study is terminated early or the last participant is lost to follow-up.

#### 6.6.4 **Definition of Study Discontinuation**

Celerion reserves the right to terminate the study in the interest of participant welfare.

The Sponsor reserves the right to suspend or terminate the study at any time, for any reason.

#### 6.6.5 Criteria for Premature Termination or Suspension of the Study

The study will be completed as planned unless one or more of the following criteria are satisfied that require temporary suspension or early termination of the study:

- New information or other evaluation regarding the safety or efficacy of the study medication that indicates a change in the known risk/benefit profile for the product, such that the risk is no longer acceptable for participants participating in the study
- Significant violation of Good Clinical Practice (GCP) that compromises the ability to achieve the primary study objectives or compromises participant safety.

#### Criteria for Premature Termination or Suspension of a Site 6.6.6

#### 6.6.6.1 Criteria for Premature Termination or Suspension

A study site may be terminated prematurely or suspended if the site (including the Investigator) is found in significant violation of GCP, the study protocol, or contractual agreement; if the site (including the Investigator) is unable to ensure adequate performance of the study; or as otherwise permitted by the contractual agreement.

#### 6.6.6.2 Procedures for Premature Termination or Suspension

In the event that the sponsor, an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), or a regulatory authority elects to terminate or suspend the participation of an investigational site, a study-specific procedure for early termination or suspension will be provided by the sponsor; the procedure will be followed by applicable investigational site(s) during the course of termination or study suspension.

# SELECTION AND DISCONTINUATION/WITHDRAWAL OF PARTICIPANTS

#### **Inclusion Criteria**

Participants must fulfill the following inclusion criteria before the first dose to be eligible for participation in the study:

- 1. Healthy, adult, male or female of non-childbearing potential (Appendix D), 18 55 years of age, inclusive, at screening.
- 2. Male participant agrees to comply with any applicable contraceptive requirements of the protocol as detailed in Appendix D.

- 3. BMI  $\geq$  18.0 and  $\leq$  32.0 kg/m<sup>2</sup> at screening.
- 4. Continuous non-smoker who has not used nicotine-containing products for at least 90 days prior to the first dosing.
- 5. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
  - Supine BP is  $\geq$ 90/40 mmHg and  $\leq$ 140/90 mmHg at screening;
  - Supine HR is  $\ge$ 45 bpm and  $\le$ 100 bpm at screening;
  - QTcF is ≤450 msec (males) or ≤470 msec (females) and ECG findings considered normal or not clinically significant by the Investigator or designee at screening;
  - Estimated creatinine clearance ≥80 mL/min at screening.
  - Liver function tests including ALT and AST  $\leq 1.5$  X the ULN at screening and check-in.
- 6. Able to swallow multiple tablets/capsules.
- 7. Understands the study procedures in the ICF, and be willing and able to comply with the protocol.

#### 7.2 Exclusion Criteria

Participants must not be enrolled in the study if they meet any of the following criteria before the first dose of study drug:

- 1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
- 2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
- 3. History or presence of gastritis, gastrointestinal tract, gastric bypass surgery, or hepatic disorder or other clinical condition which, in the opinion of the Investigator or designee, may affect the absorption, distribution, metabolism, or elimination of study drugs.
- 4. History or presence of cataracts or other clinically significant vision disturbances.
- 5. History or presence of epilepsy, seizure, or convulsion, tremor or related symptoms.
- 6. History of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
- 7. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
- 8. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.

- 11. Female participants with a positive pregnancy test at screening or check-in or who is lactating.

  12. Positive urine drug or alcohol results at screening or check-in or who is lactating. 9. Any positive responses on the C-SSRS that in the clinical judgment of the Investigator has a

- 14. Unable to refrain from or anticipates the use of:
  - Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to first dosing.
- 15. History of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to the following: beer [354 mL/12 oz], wine [118 mL/4 oz], or distilled spirits [29.5 mL/1 oz] per day).
- 16. The participant consumes excessive amounts, defined as greater than 4 servings (1 serving is approximately equivalent to 120 mg of caffeine), of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
- 17. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
- 18. Donation of blood or significant blood loss within 56 days prior to the first dosing.
- 19. Plasma donation within 7 days prior to the first dosing.
- 20. Participation in another clinical study within 30 days or 5 half-lives prior to the first dosing. The 30-days window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

# **Excluded Medications, Supplements, Dietary Products**

Concomitant medications will be prohibited as listed in the exclusion criteria in Section 7.2 and throughout the study, including the follow-up period. After the first dose, ibuprofen (up to 1.2 g per 24 hour period) may be administered at the discretion of the Investigator or designee. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to the first dosing.

atlined in and the property of the applicable terms of

| Table 7.a E | Excluded Medications, | Supplements, and | <b>Dietary Products</b> |
|---|---|---|---|
|---|---|---|---|

| | Between Screening and First Dosing (Days - | After First Dosing (Day 1) to |
|---|---|---|
| Category | 28 to predose [Day 1]) | Follow-Up |
| Alcohol | Prohibited from 48 hours prior to first dosing | Prohibited from first dosing until the end of PK collection |
| Xanthine and/or caffeine | Prohibited from 24 hours prior to first dosing <sup>a</sup> | Prohibited from first dosing until the end of PK collection <sup>a</sup> |
| Medications | See Sections 7.1 and 7.2 | See Sections 7.1 and 7.2 |
| Nicotine- and tobacco-<br>containing and/or cannabis<br>products | Prohibited from 90 days prior to first dosing | Prohibited from first dosing until the follow-up visit. |
| Food substance | | |
| Grapefruit/Seville orange | Prohibited from 14 days prior to first dosing | Prohibited from first dosing until the end of PK collection |
| Other fruit juice | Prohibited from 12 hours prior to first dosing | Prohibited from first dosing until the end of PK collection |
| Vegetables from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard), and charbroiled meats | Prohibited from 7 days prior to first dosing | Prohibited from first dosing until<br>the end of PK collection |
| Processed and grilled meat<br>consumption including but<br>not limited to sausages,<br>salami, pork flank (spiced<br>and boiled) and ham | COMMercial | Prohibited from first dosing until the end of PK collection |

(a) small amounts of caffeine derived from normal foodstuffs eg, 250 mL/8 oz/1 cup decaffeinated coffee or other decaffeinated beverage, per day, with the exception of espresso; 45 g/1.5 oz chocolate bar, per day, would not be considered a deviation to this restriction.

# 7.4 Diet, Fluid, Activity

# 7.4.1 Diet and Fluid

Water (except water provided with each dosing) will be restricted 1 hour prior to and 1 hour after each dosing, but will be allowed ad libitum at all other times. Other fluids may be given as part of meals and snacks but will be restricted at all other times throughout the confinement period.

Participants will fast overnight for at least 10 hours prior to each soticlestat dosing and at least 8 hours prior to each rifampin dosing. Participants will continue the fast for at least 4 hours on all dosing days. For limiting nitrosamine exposure from food, processed and grilled meat consumption including but not limited to sausages, salami, pork flank (spiced and boiled) and ham will be excluded from first dosing until the end of PK collection.

When confined, standard meals and snacks will be provided at appropriate times, except when they are required to fast. When confined in the CRU, participants will be required to fast from all food and drink except water between meals and snacks.

Each meal and/or snack served at the CRU will be standardized and will be similar in caloric content and composition and will be taken at approximately the same time in each period.

# 7.4.2 Activity

Participants will remain seated for the first 4 hours post soticlestat dose, except when they are supine or semi reclined for study procedures. Participants will then resume normal activity.

However, should AEs occur at any time, participants may be placed in an appropriate position or will be permitted to lie down on their right side. During the first 4 hours postdose, participants may be allowed to rise for brief periods under supervision (eg, in order to use the toilet facilities).

Participants will be instructed to refrain from strenuous physical activity which could cause muscle aches or injury, including contact sports at any time from screening until completion of the study.

# 7.5 Criteria for Discontinuation or Withdrawal of a Participant

1. Pretreatment event (PTE) or AE: The participant has experienced a PTE or AE that requires early termination because continued participation imposes an unacceptable risk to the participant's health or the participant is unwilling to continue because of the PTE or AE.

# <u>Liver Function Test (LFT) Abnormalities:</u>

Study drug should be discontinued immediately with appropriate clinical follow-up (including repeat laboratory tests, until a participant's laboratory profile has returned to normal/baseline status, see Section 9.2.9), if the following circumstances occur at any time during study drug treatment:

- ALT or AST >8 × ULN, or
- ALT or  $\overrightarrow{AST} > 5 \times ULN$  and persists for more than 2 weeks, or
- ALT or AST >3 × ULN in conjunction with elevated total bilirubin >2 × ULN or international normalized ratio (INR) >1.5, or
- ALT or AST >3 × ULN with appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (>5%).

# QTcF interval:

Study drug should be discontinued immediately with appropriate clinical follow-up if a QTcF interval >500 msec or if there is an increase of QTcF >60 mecs above screening/baseline detected by ECG and confirmed with a repeat ECG. Appropriate clinical follow-up includes a repeat ECG.

- 2. Significant protocol deviation: The discovery post-enrollment that the participant failed to meet protocol entry criteria or did not adhere to protocol requirements, and continued participation poses an unacceptable risk to the participant's health.
- 3. Lost to follow-up: Attempts to contact the participants were unsuccessful. Attempts to contact the participant must be documented in the participant's source documents.
- 4. Voluntary withdrawal: The participant (or participant's legally acceptable representative) wishes to withdraw from the study. The reason for withdrawal, if provided, should be recorded in the CRF.

Note: All attempts should be made to determine the underlying reason for the withdrawal and, where possible, the primary underlying reason should be recorded (ie, withdrawal due to an AE should not be recorded in the "voluntary withdrawal" category). If a participant chooses to withdraw from study participation due to personal concerns related to the COVID-19 pandemic (other than a COVID-19-related AE), this should be specified as the reason for participant withdrawal in the CRF.

- 5. Study termination: The Sponsor, IRB/ IEC, or regulatory agency terminates the study.
- 6. Pregnancy: as described in Appendix D.
- 7. Participants may be withdrawn from the study by the Investigator or designee for the following reasons:
  - Difficulties in blood collection.
  - Positive urine drug or alcohol test.
- 8. Other. The specific reasons for discontinuation should be entered into the CRF including unavoidable circumstances such as the COVID-19 pandemic. Participants may be withdrawn from the study at any time at the discretion of the Investigator or Sponsor for safety reasons which should be entered into the CRFs.

# 7.6 Procedures for Discontinuation or Withdrawal of a Participant

The Investigator may discontinue a participant's study participation at any time during the study when the participant meets the study termination criteria described in Section 7.5. In addition, a participant may discontinue his or her participation without giving a reason at any time during the study. Should a participant's participation be discontinued, the primary criterion for termination must be recorded by the Investigator. In addition, efforts should be made to perform all procedures scheduled for the end-of-study or early termination as described in Section 3.0.

## 7.7 Participant Replacement

Replacement of discontinued or withdrawn participants due to any reason will be assessed on a case by case basis by the Sponsor and Investigator to ensure a minimum of 12 PK-evaluable participants complete the study.

#### 8.0 CLINICAL STUDY MATERIAL MANAGEMENT

# 8.1 Clinical Study Drug

## **Investigational Medicinal Product**

Product Name: Soticlestat (TAK-935)

Strength: 100 mg

Dose: 300 mg (3 x 100 mg strength)

Dosage Form/Formulation: T4 immediate release tablet

Dosing regimen: Single dose

Route of Administration: Oral

**Interacting Drug** 

Product Name: Rifampin

Strength: 300 mg

Dose: 600 mg (2 x 300 mg strength)

Dosage Form/Formulation: Capsule

Dosing regimen: Multiple dose (QD)

Route of Administration: Oral

Preference for generic or brand name. Brand name or generic.

# 8.1.1 Clinical Study Drug Labeling

Study drug containers will be affixed with a clinical label in accordance with local regulatory requirements.

# 8.1.2 Clinical Study Drug Inventory and Storage

The Sponsor will supply sufficient quantities of soticlestat to allow completion of this study. Celerion will supply sufficient quantities of rifampin to allow completion of this study.

For each study medication (ie, soticlestat and rifampin), the same lot number will be used throughout the study. The lot numbers and expiration dates (where available) of the study drugs supplied will be recorded in the final report. Study drugs will be stored according to the product labels provided with the product.

Records will be made of the receipt, preparation, dispensing, and final disposition of the study drugs supplied.

# 8.1.3 Clinical Study Drug Blinding

This is an open-label study.

#### 8.1.4 **Randomization Code Creation and Storage**

Not applicable.

#### 8.1.5 Clinical Study Blind Maintenance/Unblinding Procedure

Not applicable.

#### **Accountability and Destruction of Sponsor-Supplied Drugs** 8.1.6

Records will be made of the receipt and dispensing of the study drugs supplied. At the conclusion of the study, any unused soticlestat will be retained by Celerion, returned to the Sponsor or designee, or destroyed, as per Sponsor instructions. Any remaining supplies that were purchased by Celerion will be destroyed, if appropriate. If no supplies remain, this fact will be documented in the pharmacy product accountability records. and Subject

#### 9.0 STUDY PROCEDURES

#### 9.1 Administrative Procedures

#### 9.1.1 **Informed Consent Procedure**

The purpose of the study, the procedures to be carried out and the potential hazards will be described to the participant in non-technical terms. Participants will be required to read, sign, and date an ICF summarizing the discussion prior to screening, and will be assured that they may withdraw from the study at any time without jeopardizing their medical care.

Participants will be given a copy of their signed ICF.

#### Assignment of Screening Numbers 9.1.1.1

Each participant will be assigned a unique identification number upon screening. Participants who complete the study screening assessments and meet all the eligibility criteria will be assigned a unique identification number at the time of dosing in Period 1, different from the screening number.

If replacement participants are used, the replacement participant number will be 100 more than the original participant's identification number (eg. Participant No. 101 will assigned to the replacement of Participant No. 1).

#### 9.1.0.2 Study Drug Assignment

All participants will receive the treatments as detailed in Section 9.2.6.

#### 9.1.2 **Inclusion and Exclusion**

Please refer to Section 7.1 and Section 7.2.

## 9.1.3 Medical History/Demography

Medical history and demographic data, including name, sex, age, race, ethnicity, and history of tobacco use will be recorded.

#### 9.1.4 Concomitant Medications

Concomitant medications will be prohibited as listed in Section 7.3. All medications taken by participants during the course of the study will be recorded.

#### 9.2 Clinical Procedures and Assessments

The Schedule of Study Procedures (Section 3.0) summarizes the clinical procedures to be performed at each visit. Individual clinical procedures are described in detail below. Additional evaluations/testing may be deemed necessary by the Investigator or designee and/or the Sponsor for reasons related to participant safety.

For this study, collection of blood for soticlestat

the critical parameter and needs to be collected as close to the exact time point as possible. All other procedures should be completed as close to the prescribed/scheduled time as possible, but can be performed prior to or after the prescribed/scheduled time.

Any nonscheduled procedures required for urgent evaluation of safety concerns take precedence over all routine scheduled procedures.

## 9.2.1 Physical Exam

A full and abbreviated physical examination will be performed as outlined in the Schedule of Study Procedures (Section 3.0).

An abbreviated physical examination will include at the minimum, examination of respiratory, cardiovascular, and gastrointestinal systems, with the option for further examination of additional systems as necessary based on reported symptoms/AEs.

Symptom-driven physical examinations may be performed at other times, if deemed necessary by the Investigator or designee.

# 9.2.2 Height and Weight

Body height (cm) and weight (kg) will be reported as outlined in the Schedule of Study Procedures (Section 3.0).

#### 9.2.3 BMI

BMI will be calculated based on the height and weight measured at screening.

## 9.2.4 Vital Signs

Single measurements of temperature, respiratory rate, blood pressure and pulse rate, will be measured as outlined in the Schedule of Study Procedures (Section 3.0). Additional vital signs may be taken at any other times, if deemed necessary.

Blood pressure and pulse rate measurements will be performed with participants in a supine position (5 minutes).

Vital signs will be measured within 24 hours prior to Day 1 dosing of Period 1 for the predose time point. At all other predose time points, vital signs will be measured within 2 hours prior to dosing. When scheduled postdose, vital signs will be performed within approximately 15 minutes of the scheduled time point.

## 9.2.5 12-Lead ECG

Single 12-lead ECGs will be performed as outlined in the Schedule of Study Procedures (Section 3.0). Additional ECGs may be taken at any other times, if deemed necessary by the Investigator or designee.

ECGs will be performed with participants in a supine position (5 minutes). All ECG tracings will be reviewed by the Investigator or designee.

ECGs will be measured within 24 hours prior to Day 1 dosing of Period 1 for the predose time point. At all other predose time points, ECGs will be collected within 2 hours prior to dosing. When scheduled postdose, ECGs will be performed within approximately 20 minutes of the scheduled time point.

## 9.2.6 Study Drug Administration

Study drugs and study drug formulations will be provided as described in Section 8.1.

Dose regimens for study drugs are described in Table 2.b.

After initial morning dosing on Day 1 of Period 2, each subsequent study drug dose will be administered within  $\pm$  1 hour of dosing time established on Day 1 of Period 2.

The pharmacy at the CRU will provide each dose in individual unit dose containers for each participant, as appropriate.

Study drugs will be administered with approximately 240 mL of water.

Additional information regarding drug preparation and administration may be provided in a separate document.

Participants will be instructed not to crush, split, or chew the tablets and/or capsules.

The exact clock time of dosing will be recorded.

A qualified designee will be responsible for monitoring the administration of the assigned doses. A mouth check will be performed by the qualified designee to ensure that the participants have swallowed the study drug(s). Once a participant has finished the dosing water, the qualified

designee will use a flashlight and a tongue depressor to check the participant's mouth. Participants' hands will also be verified to ensure that the study drug(s) was ingested.

#### 9.2.7 C-SSRS

Suicidal ideation will be assessed using the C-SSRS at the times stipulated in the Schedule of Study Procedures (Section 3.0) for each study part. Two versions of the C-SSRS will be used in this study: the Screening/Baseline C-SSRS Lifetime and the Since-Last-Visit C-SSRS. It is recommended that the same staff be used to administer the scale to the participant at all time points when C-SSRS is scheduled. Any suicidal ideation or suicidal behavior during the trial periods detected by the C-SSRS will be recorded as an AE. The Investigator will ensure that any suicidal ideation or behavior is medically addressed, including assessment and treatment by qualified medical personnel.

## 9.2.8 **AE Monitoring**

Participants will be monitored throughout the study for adverse reactions to the study drugs and/or procedures as described in Section 10.0.

# 9.2.9 Laboratory Procedures and Assessments

All tests listed below will be performed as outlined in the Schedule of Study Procedures (Section 3.0). In addition, laboratory safety tests may be performed at various unscheduled time points, if deemed necessary by the Investigator or designee.

## 9.2.9.1 Clinical Laboratory Tests

#### <u>Hematology</u>

Hematology will consist of the following tests:

| Hemoglobin | Red blood cell count |
|---|---|
| Hematocrit | Platelet count |
| Erythrocytes | Mean platelet volume |
| Total and differential leukocyte count | Immune cell count (neutrophils, lymphocytes, |
| | monocytes, eosinophils, basophils) |

#### <u>Coagulation</u>

Coagulation test will be conducted as outlined in the Schedule of Study Procedures (Section 3.0). Coagulation test will consist of the following tests:

| Activated partial thromboplastin time |
|---------------------------------------------------|
| Prothrombin time / International normalized ratio |

## **Chemistry**

Serum chemistry tests will be performed after at least an 8-hour fast; however, in case of dropouts or rechecks, participants may not have fasted for 8 hours prior to when the serum chemistry sample is taken.

Chemistry evaluations will consist of the following standard chemistry panel:

| Blood Urea Nitrogen | Albumin |
|---|---|
| Bilirubin (total, direct and indirect) | Sodium |
| Alkaline phosphatase (ALP) | Potassium |
| Aspartate aminotransferase (AST) | Chloride |
| Alanine aminotransferase (ALT) | Glucose |
| Calcium | Creatinine ** |
| Carbon dioxide | Phosphate |
| Protein (total) | Alpha1-acidic glycoprotein (AGP) (screening only) |
| Gamma-glutamyl transferase (GGT) | Magnesium |
| Urea | 29 |

<sup>\*</sup> At screening, creatinine clearance will be calculated using the Cockcroft-Gault formula.

## <u>Urinalysis</u>

Urinalysis will consist of the following tests:

| рН | 1)3 | Bilirubin |
|------------------|------------------|----------------------|
| Specific gravity | :0 | Blood * |
| Protein * | ar <sub>CO</sub> | Nitrite * |
| Glucose | in | Urobilinogen |
| Ketones | | Leukocyte esterase * |
| Erythrocytes | Ö | Creatinine |
| Calcium | 1011 | |

<sup>\*</sup> If urinalysis is positive for protein, blood, nitrite and/or leukocyte esterase, a microscopic examination (for red blood cells, white blood cells, bacteria, casts, and epithelial cells) will be performed.
## 9.2.9.1.1 <u>Other</u>

| HIV test | Urine drug screen |
|---|---|
| HBsAg | - Opiates (includes morphine, heroin (diacetylmorphine), |
| HCV (if antibody positive, confirm RNA negative) | codeine, 6-acetylmorphine, dihydrocodeine, hydrocodone, thebaine, and, hydromorphone) |
| Urine alcohol screen | - Amphetamines |
| Serum pregnancy test (for females only) | |
| FSH (for females only) | Benzodiazepines |
| COVID-19 (SARS-CoV-2 polymerase chain reaction test or equivalent) | <ul> <li>Barbiturates</li> <li>Benzodiazepines</li> <li>Cocaine</li> <li>Cannabinoids</li> </ul> |
| | - Buprenorphine/metabolite |
| | - MDMA(3,4-methylenedioxy-methamphetamine) |
| | - Methadone/metabolite |
| | - Oxycodone/oxymorphone |
| | - Phencyclidine |

### 9.3 Pharmacokinetic Samples

Samples for assessment of soticlestat as delineated in Table 9.a.

) will be collected

Instructions for sample collection, processing, and shipping will be provided in separate documents.

Primary specimen collection parameters are provided in Table 9.a.

**Table 9.a** Primary Specimen Collections

| Specimen Name | Primary<br>Specimen | Primary<br>Specimen<br>Derivative | Description of Intended Use | Sample<br>Collection |
|---|---|---|---|---|
| Plasma sample for soticlestat | Blood | Plasma | Plasma sample for PK analysis | Mandatory |

## 9.3.1 **Pharmacokinetic Measurements**

Samples from all participants will be assayed even if the participants do not complete the study. Samples for determination of plasma soticlestat will be analyzed using validated bioanalytical methods.

PK parameters of soticlestat will be calculated from the individual concentration-time profiles from all evaluable participants using noncompartmental analysis methods. Actual sampling times, rather than scheduled sampling times, will be used in all computations involving sampling times.

#### 9.3.1.1 Plasma for PK Measurements

The following PK parameters will be calculated from plasma concentrations of soticlestat unless otherwise specified:

AUC<sub>last</sub>: The area under the concentration-time curve, from time 0 to the last

insofuse quantifiable concentration, as calculated by the linear-log trapezoidal

method.

The area under the concentration-time curve, from time 0 extrapolated to  $AUC_{\infty}$ :

infinity. AUC $_{\infty}$  is calculated as AUC<sub>last</sub> plus the ratio of the last measurable

blood concentration to the elimination rate constant.

Percent of  $AUC_{\infty}$  extrapolated, represented as  $(1 - AUC_{last}/AUC_{\infty})*100$ . AUC<sub>extrap</sub>%:

CL/F: Apparent total plasma clearance after oral (extravascular) administration,

calculated as Dose/AUC<sub>∞</sub> (soticlestat only).

Maximum observed concentration. C<sub>max</sub>:

Time to reach C<sub>max</sub>. If the maximum value occurs at more than one time t<sub>max</sub>:

point, t<sub>max</sub> is defined as the first time point with this value.

Terminal disposition phase rate constant.  $\lambda_z$ 

Terminal disposition phase half-life will be calculated as  $0.693/\lambda_z$ .  $t^{1/2}$ :

> Where  $\lambda_z$  is the apparent first order terminal disposition phase rate constant calculated from a semilog plot of the plasma concentration versus time curve. The parameter will be calculated by linear least-squares- regression analysis using the maximum number of points in the terminal log-linear

phase (eg, three or more non-zero plasma concentrations).

Apparent volume of distribution during the terminal disposition phase after  $V_z/F$ :

oral (extravascular) administration, calculated as Dose/(AUC $_{\infty}$ x  $\lambda_z$ )

(soticlestat only).

No value for  $\lambda_z$ ,  $AUC_{\infty}$ ,  $AUC_{\text{extrap}}$ %, CL/F,  $V_z/F$ ,  $\lambda z$ , or  $t\frac{1}{2}$  will be reported for cases that do not exhibit a terminal log-linear phase in the concentration versus time profile.

No PK parameters will be calculated for participants with detectable concentrations at 2 or fewer consecutive time points.

Individual and mean plasma concentration-curves (both linear and log-linear) will be included in the final report.

Additional PK parameters may be estimated as appropriate.

#### 9.3.2 **Biomarker Measurements**

Not applicable.

#### 9.3.3 PGx Measurements

Not applicable.

#### 9.3.4 Confinement

Participants will be housed on Day -1 of Period 1, at the time indicated by the CRU, until after the last blood draw and/or study procedures on Day 14 of Period 2. Participants may be asked to check-in to the CRU earlier to undergo additional COVID 19 precaution procedures or testing not related to study protocol, as per CRU requirements.

At all times, a participant may be required to remain at the CRU for longer at the discretion of the Investigator or designee.

The CRU will contact all participants (including participants who terminate the study early)  $15 \pm 2$  days after the last soticlestat administration to determine if any AEs have occurred since the last study visit. If clinically significant findings are observed upon discharge, participants may return to the CRU for re-evaluation per Investigator's discretion.

#### 10.0 ADVERSE EVENTS

#### 10.1 Definitions and Elements of AEs

An AE is defined as any untoward medical occurrence in a clinical investigation participant who has signed informed consent to participate in a study; it does not necessarily have to have a causal relationship with the treatment.

An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.

An untoward finding generally may:

- Indicate a new diagnosis or unexpected worsening of a preexisting condition. (Intermittent events for pre-existing conditions or underlying disease should not be considered AEs.)
- Necessitate therapeutic intervention.
- Require an invasive diagnostic procedure.
- Require discontinuation or a change in dose of study medication or a concomitant medication.
- Be considered unfavorable by the investigator for any reason.

Diagnoses versus signs and symptoms:

• Each event should be recorded to represent a single diagnosis. Accompanying signs (including abnormal laboratory values or ECG findings) or symptoms should NOT be recorded as additional AEs. If a diagnosis is unknown, sign(s) or symptom(s) should be recorded appropriately as an AE(s).

#### Laboratory values and ECG findings:

- Changes in laboratory values or ECG parameters maybe considered AEs if they are judged to be clinically significant (ie, if some action or intervention is required or if the investigator judges the change to be beyond the range of normal physiologic fluctuation). A laboratory retest and/or continued monitoring of an abnormal value are not considered an intervention. In addition, repeated or additional noninvasive testing for verification, evaluation or monitoring of an abnormality is not considered an intervention.
- If abnormal laboratory values or ECG findings are the result of pathology for which there is an overall diagnosis (eg, increased creatinine in renal failure), the diagnosis only should be reported appropriately as an AE.

### Pre-existing conditions:

- A pre-existing condition (present at the time of signing of informed consent) is considered a concurrent medical history condition and should NOT be recorded as an AE. A baseline evaluation (eg, laboratory test, ECG, X-ray, etc) should NOT be recorded as an AE unless related to a study procedure. However, if the participant experiences a worsening or complication of such a concurrent medical history condition, the worsening or complication should be recorded appropriately as an AE (worsening or complication occurs after informed consent is signed). Investigators should ensure that the event term recorded captures the change in the condition (eg, "worsening of...").
- If a participant has a pre-existing episodic condition (eg, asthma, epilepsy), any occurrence of an episode should only be captured as an AE if the episodes become more frequent, serious, or severe in nature, that is, investigators should ensure that the AE term recorded captures the change from Baseline in the condition (eg "worsening of...").
- If a participant has a degenerative concurrent condition (eg, cataracts, rheumatoid arthritis), worsening of the condition should only be captured as an AE if occurring to a greater extent to that which would be expected. Again, investigators should ensure that the AE term recorded captures the change in the condition (eg, "worsening of...").

# Worsening of AEs.

• If the participant experiences a worsening or complication of an AE after the first administration of study medication or after any change in study medication, the worsening or complication should be recorded as a new AE. Investigators should ensure that the AE term recorded captures the change in the condition (eg, "worsening of...").

# Changes in severity of AEs:

• If the participant experiences a change in the severity of an AE that is not associated with a change in study medication, the event should be captured once with the maximum severity recorded.

#### Preplanned surgeries or procedures:

Preplanned procedures (surgeries or therapies) that were scheduled prior to signing of
informed consent are not considered AEs. However, if a preplanned procedure is performed
early (eg, as an emergency) due to a worsening of the pre-existing condition, the worsening
of the condition should be captured appropriately as an AE. Complications resulting from
any planned surgery should be reported as AEs.

#### Elective surgeries or procedures:

• Elective procedures performed where there is no change in the participant's medical condition should not be recorded as AEs but should be documented in the participant's source documents. Complications resulting from an elective surgery should be reported as AEs.

#### Overdose:

- An overdose is defined as a known deliberate or accidental administration of investigational
  drug, to or by a study participant, at a dose above that which is assigned to that individual
  participant according to the study protocol. It is up to the investigator or the reporting
  physician to decide whether a dose is to be considered an overdose, in consultation with the
  Sponsor.
- All cases of overdose (with or without associated AEs) will be documented on an Overdose page of the (e)CRF, in order to capture this important safety information consistently in the database. AEs associated with an overdose will be documented on AE CRF(s) according to Section 10.0.
- Serious adverse events (SAEs) of overdose should be reported according to the procedure outlined in Section 10.2.8.
- In the event of drug overdose, the participant should be treated symptomatically.

#### 10.1.1 SAEs

An SAE is defined as any untoward medical occurrence that at any dose:

- 1. Results in DEATH.
- 2. Is LIFE THREATENING.
  - The term "life threatening" refers to an event in which the participant was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.
- 3. Requires inpatient HOSPITALIZATION or prolongation of existing hospitalization.
- 4. Results in persistent or significant DISABILITY/INCAPACITY.
- 5. Is a CONGENITAL ANOMALY/BIRTH DEFECT.
- 6. Is an IMPORTANT MEDICAL EVENT that satisfies any of the following:

- May require intervention to prevent items 1 through 5 above.

Table 10.a

| • May require intervention to prevent items 1 through 5 above. | |
|---|---|
| <ul> <li>May require intervention to prevent items 1 through 5 above.</li> <li>May expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization.</li> </ul> | |
| • Includes any event or synonym of (Table 10.a). | described in the Takeda Medically Significant AE List |
| Table 10.a Takeda Medically Significant AE List | |
| | Term |
| Acute respiratory failure/acute respiratory | Hepatic necrosis |
| distress syndrome | Acute liver failure Anaphylactic shock |
| Torsade de pointes / ventricular fibrillation / | Anaphylactic shock |
| ventricular tachycardia | Acute renal failure |
| Malignant hypertension | Pulmonary hypertension |
| Convulsive seizures | Pulmonary fibrosis |
| Agranulocytosis | Confirmed or suspected endotoxin shock |
| Aplastic anemia | Confirmed or suspected transmission of infectious agent |
| Toxic epidermal necrolysis/ | by a medicinal product |
| Stevens-Johnson syndrome | Neuroleptic malignant syndrome / malignant hyperthermia |
| COVID-19 pneumonia | Spontaneous abortion / stillbirth and fetal death |
| COVID-19-related disease | 150 |

Abbreviations: COVID-19 = Coronavirus disease-2019

AEs that fulfill 1 or more of the serious criteria above are to be considered SAEs and should be reported and followed up in the same manner (see Sections 10.1 and 10.1.1).

#### 10.1.2 Special Interest AEs

There are no AEs of Special Interest for this study.

#### 10.2 AE Procedures

#### Assigning Severity/Intensity of AEs 10.2.1

The different categories of severity/intensity are:

Mild: An AE that is usually transient and may require only minimal treatment or

therapeutic intervention. The event does not generally interfere with usual

activities of daily living.

Moderate: An AE that is usually alleviated with additional specific therapeutic

> intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research

participant.

Severe:

An AE that interrupts usual activities of daily living, or significantly affects

Assigning Causality of AEs

The relationship of each AE to study medication(s) will be assessed using the following categories:

Related:

An AE that follows a reasonable termon drug (including):

relationship is at least a reasonable possibility, ie, the relationship cannot be ruled out, although factors other than the drug, such as underlying diseases. complications, concomitant drugs and concurrent treatments, may also be

responsible.

Not Related: An AE that does not follow a reasonable temporal sequence from

> administration of a drug and/or that can reasonably be explained by other factors, such as underlying diseases, complications, concomitant medications

and concurrent treatments.

In addition, relationship (causality) to COVID-19 should be determined for all PTEs and AEs. The relationship should be assessed as related if the investigator considers that there is reasonable possibility that an event is due to COVID-19. Otherwise, the relationship should be assessed as not related.

Similarly, relationship (causality) to COVID-19 vaccines should be determined for all PTEs and AEs. The relationship should be assessed as related if the investigator considers that there is reasonable possibility that an event is due to COVID-19 vaccines. Otherwise, the relationship should be assessed as not related. If the AE has relationship to vaccination, specific verbatim term should be used, eg. post-vaccination fever, vaccination site burning.

In addition, if the causality assessment done by the investigator determines that the event or events (PTEs or AEs) are related or possible related to COVID-19 or the COVID-19 vaccine, the events should be assessed as not related to the investigational product. If the AE is related to COVID-19 vaccination, specific verbatim term(s) should be used, eg, post-vaccination fever, vaccination site burning.

#### 10.2.3 **Start Date**

The start date of the AE is the date that the first signs/symptoms were noted by the participant and/or investigator.

#### 10.2.4 **End Date**

The end date of the AE is the date at which the participant recovered, the event resolved but with sequelae or the participant died.

#### **10.2.5** Pattern of Adverse Event (Frequency)

Episodic AEs (eg, headache) or those which occur repeatedly over a period of consecutive days are intermittent. All other events are continuous.

#### **10.2.6** Action Taken With Study Treatment

- Drug withdrawn a study medication is stopped due to the particular AE.
- Dose not changed the particular AE did not require stopping a study medication.
- Unknown only to be used if it has not been possible to determine what action has been taken.
- Not applicable a study medication was stopped for a reason other than the particular AE eg, the study has been terminated, the participant died, dosing with study medication had not yet started or dosing with study medication was already stopped before the onset of the AE.
- Drug interrupted the dose was interrupted due to the particular AE.

#### **10.2.7 Outcome**

- Recovered/resolved participant returned to first assessment status with respect to the AE.
- Recovering/resolving the intensity is lowered by one or more stages: the diagnosis has or signs/symptoms have almost disappeared, the abnormal laboratory value improved, but has not returned to the normal range or to the baseline value; the participant died from a cause other than the particular AE with the condition remaining "recovering/resolving."
- Not recovered/not resolved there is no change in the diagnosis, signs or symptoms; the intensity of the diagnosis, signs/symptoms or laboratory value on the last day of the observed study period has become worse than when it started; is an irreversible congenital anomaly; the participant died from another cause with the particular AE state remaining "Not recovered/not resolved."
- Recovered/Resolved with sequelae the participant recovered from an acute AE but was left with permanent/significant impairment (eg, recovered from a cardiovascular accident but with some persisting paresis).
- Fatal an AE that is considered as the cause of death.
- Unknown the course of the AE cannot be followed up due to hospital change or residence change at the end of the participant's participation in the study.

### 10.2.8 Collection and Reporting of AEs, SAEs, Special Interest AEs, and Abnormal LFTs

#### 10.2.8.1 Collection Period

Collection of AEs (ie, AEs, SAEs, Special Interest AEs, and Abnormal LFTs) will commence at the time the participant signs the informed consent. Routine collection of AEs will continue until

the follow-up contact 15 ( $\pm$  2) days after last dose of soticlestat. For participants who discontinue prior to the administration of study medication, AEs will be followed until the participant discontinues study participation.

### 10.2.8.2 Reporting AEs

At each study visit, the investigator will assess whether any subjective AEs have occurred. A neutral question, such as "How have you been feeling since your last visit?" may be asked. Participants may report AEs occurring at any other time during the study. Participants experiencing an SAE prior to the first exposure to investigational product must be monitored until the symptoms subside and any clinically relevant changes in laboratory values have returned to Baseline or there is a satisfactory explanation for the change. Nonserious AEs that begin prior to the first exposure to investigational product, related or unrelated to the study procedure, need not be followed-up for the purposes of the protocol.

All participants experiencing AEs, whether considered associated with the use of the study medication or not, must be monitored until the symptoms subside and any clinically relevant changes in laboratory values have returned to Baseline or until there is a satisfactory explanation for the changes observed. All AEs will be documented in the AE page of the CRF, whether or not the investigator concludes that the event is related to the drug treatment. The following information will be documented for each event:

- Event term.
- Start and end date and time.
- Pattern of AE (frequency).
- Severity/Intensity.
- Causality (Investigator's opinion of the causal relationship between the event and administration of study drug[s]).
- Relationship to COVID-19.
- Relationship to COVID-19 vaccine.
- Action taken with study drug.
- Outcome of event.
- Seriousness.

# 10.2.8.3 Reporting SAEs

When an SAE occurs through the AE collection period it should be reported according to the procedure outlined below:

A Takeda SAE form must be completed, in English and signed by the investigator immediately or within 24 hours of first onset or notification of the event. The information should be completed as fully as possible but contain, at a minimum:

- A short description of the event and the reason why the event is categorized as serious.
- Participant identification number.
- Investigator's name.
- Name of the study medication(s).
- Causality assessment.

The SAE form should be transmitted within 24 hours to the attention of the contact listed in Appendix 14.1.1.

Any SAE spontaneously reported to the investigator following the AE collection period should be reported to the Sponsor if considered related to study participation.

Reporting of SAEs that begin before first administration of investigational product will follow the same procedure for SAEs occurring on treatment.

## 10.2.8.3.1 <u>SAE Follow-Up</u>

If information is not available at the time of the first report becomes available at a later date, the investigator should complete a follow-up SAE form or provide other written documentation and fax it immediately within 24 hours of receipt. Copies of any relevant data from the hospital notes (eg, ECGs, laboratory tests, discharge summary, postmortem results) should be sent to the addressee, if requested.

All SAEs should be followed up until resolution or permanent outcome of the event. The timelines and procedure for follow-up reports are the same as those for the initial report.

## 10.2.8.4 Reporting Special Interest AEs

There are no AEs of Special Interest for soticlestat.

# 10.2.8.5 Reporting of Abnormal LFTs

If a participant is noted to have ALT or AST elevated >3 ×ULN on 2 consecutive occasions, the abnormality should be recorded as an AE. In addition, an LFT Increases CRF must be completed providing additional information on relevant recent history, risk factors, clinical signs and symptoms and results of any additional diagnostic tests performed.

If a participant is noted to have ALT or AST >3 ×ULN and total bilirubin >2 ×ULN for which an alternative etiology has not been identified, the event should be recorded as an SAE and reported as per Section 10.2.8.3. The investigator must contact the Medical Monitor for discussion of the relevant participant details and possible alternative etiologies, such as acute viral hepatitis A or B or other acute liver disease. Follow-up laboratory tests as described in Section 9.2.8 must also be performed. In addition, an LFT Increases CRF must be completed and transmitted with the Takeda SAE form (as per Section 10.2.9).

## 10.2.9 Safety Reporting to Investigators, IRBs or IECs, and Regulatory Authorities

The Sponsor will be responsible for reporting all suspected unexpected serious adverse reactions (SUSARs) and any other applicable SAEs to regulatory authorities, investigators and IRBs or IECs, as applicable, in accordance with national regulations in the countries where the study is conducted. Relative to the first awareness of the event by/or further provision to the Sponsor or Sponsor's designee, SUSARs will be submitted within 7 days for fatal and life-threatening events and 15 days for other serious events, unless otherwise required by national regulations. The Sponsor will also prepare an expedited report for other safety issues where these might materially alter the current benefit-risk assessment of an investigational medicinal product or that would be sufficient to consider changes in the investigational medicinal products administration or in the overall conduct of the study. The investigational site also will forward a copy of all expedited reports to his or her IRB or IEC in accordance with national regulations.

#### 11.0 STATISTICAL METHODS

## 11.1 Statistical and Analytical Plans

Detailed methodology for summary and statistical analyses of the data collected in this study will be documented in a statistical analysis plan (SAP). This document may modify the plans outlined in the protocol; however, any major modifications of the primary endpoints definition and/or its analysis will also be reflected in a protocol amendment. Additional statistical analyses other than those described in this section may be performed if deemed appropriate.

#### 11.1.1 Analysis Sets

#### 11.1.1.1 PK Set

All participants who comply sufficiently with the protocol and display an evaluable PK profile (eg, exposure to treatment, availability of measurements and absence of major protocol violations) will be included in the PK set. More details will be provided in SAP.

# 11.1.1.2 Safety Set

All participants who received at least one dose of the study drug(s) will be included in the safety set.

# 11.1,2 Analysis of Demography and Other Baseline Characteristics

Continuous demographic data (ie, age, weight, height, and BMI) will be listed and summarized using appropriate summary statistics. Categorical demographic data (ie, gender, race, and ethnicity) will also be listed and tabulated.

#### 11.1.3 PK Analysis

Statistical analysis of PK data will be based on the PK analysis data set.

Values will be reported for the plasma soticlestat concentrations for each participant. PK parameters for plasma concentrations of soticlestat will be calculated as described in Section 9.3.1.1, and outlined in the SAP.

### 11.1.3.1 Linear Mixed Effects Models

Ln-transformed  $AUC_{last}$ ,  $AUC_{\infty}$ , and  $C_{max}$  data will be analyzed using a linear mixed effects model, separately. The model will include treatment (soticlestat with and without rifampin) as a fixed-effect and participant as a random effect. The point estimates and 90% CIs for the GMRs of  $AUC_{\infty}$ ,  $AUC_{last}$ , and  $C_{max}$  for soticlestat with versus without rifampin will be calculated using the exponentiation of the point estimates of the difference between treatment regimen and the corresponding 90% CIs from the analyses on the ln-transformed  $AUC_{last}$ ,  $AUC_{\infty}$ , and  $C_{max}$ .

#### 11.1.3.2 Non-Parametric Analysis

• t<sub>max</sub> will be analyzed using nonparametric analysis for paired samples (the Wilcoxon Signed Rank Test statistic). The difference of medians (treatment effect) and the corresponding 90% CI will be estimated using the Hodges-Lehmann method and Walsh Averages. tmax will not be ln-transformed. The comparisons of interest is the same as the analysis described in Section 11.1.3.1.

#### 11.1.4 PD Analysis

Not applicable.

# 11.1.5 Safety Analysis

All safety data will be populated in the individual CRFs.

Dosing dates and times will be listed by participant.

TEAEs will be tabulated. The remaining quantitative safety data as well as the difference to baseline, when appropriate, will be summarized using the appropriate descriptive statistics.

AES will be coded using the most current version of Medical Dictionary for Regulatory Activities (MedDRA®) available at Celerion and summarized by treatment days (soticlestat alone [Period 1 Days 1 - predose Day 5]; rifampin alone [Period 2 Day 1 postdose – Day 11 predose]; and soticlestat+rifampin [Day 11 postdose to end of study]) for the number of participants reporting the TEAE and the number of TEAEs reported. A by-participant AE data listing including verbatim term, coded term, treatment, severity, and relationship to treatment will be provided.

## 11.1.5.2 Clinical Laboratory Evaluation

Clinical laboratory results will be summarized by baseline and treatment days (soticlestat alone [Period 1 Days 1 - predose Day 5]; rifampin alone [Period 2 Day 1 postdose – Day 11 predose]; and soticlestat+rifampin [Day 11 postdose to end of study]). Point of time of collection and a shift table describing out of normal range shifts will be provided.

## 11.1.5.3 *Vital Signs*

Vital signs assessments will be summarized by baseline and treatment days (soticlestat alone [Period 1 Days 1 - predose Day 5]; rifampin alone [Period 2 Day 1 postdose – Day 11 predose]; and soticlestat+rifampin [Day 11 postdose to end of study]) and point of time of collection.

## 11.1.5.4 Other Safety Parameters

Physical examination findings will be presented in the data listings.

ECGs baseline and treatment days (soticlestat alone [Period 1 Days 1 - predose Day 5]; rifampin alone [Period 2 Day 1 postdose – Day 11 predose]; and soticlestat+rifampin [Day 11 postdose to end of study]) and point of time of collection.

C-SSRS results will be summarized by point of time of collection.

Medical history, and concurrent conditions will be coded using the MedDRA® and concomitant medications will be coded using the World Health Organization (WHO) drug dictionary and will be listed by participant.

# 11.2 Interim Analysis and Criteria for Early Termination

Not applicable.

### 11.3 Determination of Sample Size

This study is not powered for hypothesis testing and is not based on any specific no-effect boundaries. The sample size is based on an estimation approach and is considered sufficient to provide a reliable estimate of the DDI magnitude.



A total of 14 participants will be dosed to ensure that 12 evaluable subjects complete the study.

#### 12.0 QUALITY CONTROL AND QUALITY ASSURANCE

#### 12.1 **Study-Site Monitoring Visits**

Msofuse Monitoring visits to the study site will be made periodically during the study to ensure that all aspects of the protocol are followed. Due to COVID-19, monitoring visits may also be conducted remotely. Source documents will be reviewed for verification of data recorded on the CRFs. Source documents are defined as original documents, data, and records. The investigator and study site guarantee access to source documents by the Sponsor or its designee contract research organisation) and by the IRB or IEC.

All aspects of the study and its documentation will be subject to review by the Sponsor or the Sponsor's designee (as long as blinding is not jeopardized), including but not limited to the Investigator's Binder, study drug, participant medical records, informed consent documentation, and review of CRFs and associated source documents. It is important that the investigator and other study personnel are available during the monitoring visits and that sufficient time is devoted to the process.

#### 12.2 **Protocol Deviations**

The investigator should not deviate from the protocol, except where necessary to eliminate an immediate hazard to study participants. Should other unexpected circumstances arise that will require deviation from protocol-specified procedures, the investigator should consult with the sponsor or designee (and IRB or IEC, as required) to determine the appropriate course of action. There will be no exemptions (a prospectively approved deviation) from the inclusion or exclusion criteria.

For COVID-19-related protocol deviations, the specific protocol deviation, the reason for the deviation, and the relationship to COVID-19 should be documented using CRU standard processes.

Significant deviations include, but are not limited to, those that involve fraud or misconduct, increase the health risk to the participant, or confound interpretation of primary study assessment.

# **Quality Assurance Audits and Regulatory Agency Inspections**

The study site also may be subject to quality assurance audits by the Sponsor or designees. In this circumstance, the Sponsor-designated auditor will contact the site in advance to arrange an auditing visit. The auditor may ask to visit the facilities where laboratory samples are collected, where the medication is stored and prepared, and any other facility used during the study. In addition, there is the possibility that this study may be inspected by regulatory agencies, including those of foreign governments (eg, the FDA, the United Kingdom Medicines and Healthcare products Regulatory Agency, the Pharmaceuticals and Medical Devices Agency of Japan). If the study site is contacted for an inspection by a regulatory body, the Sponsor should

be notified immediately. The investigator guarantees access for quality assurance auditors to all

Inis study will be conducted with the highest respect for the individual participants (ie participants) according to the protocol, the ethical principles that have their origin in the Declaration of Helsinki, and the International Conference on Harmonisation (ICH) Harmonical or regional regulatory requirements and of "Responsibilities of the Image of the are addressed through the protocol and through appendices containing requirements for informed consent and investigator responsibilities.

#### 13.1 IRB and/or IEC Approval

IRBs and IECs must be constituted according to the applicable state and federal/local requirements of each participating region. The Sponsor or designee will require documentation noting all names and titles of members who make up the respective IRB or IEC. If any member of the IRB or IEC has direct participation in this study, written notification regarding his or her abstinence from voting must also be obtained. Those Americas sites unwilling to provide names and titles of all members due to privacy and conflict of interest concerns should instead provide a Federal Wide Assurance Number or comparable number assigned by the Department of Health and Human Services.

The Sponsor or designee will supply relevant documents for submission to the respective IRB or IEC for the protocol's review and approval. This protocol, the Investigator's Brochure, a copy of the informed consent form, and, if applicable, participant recruitment materials and/or advertisements and other documents required by all applicable laws and regulations, must be submitted to a central or local IRB or IEC for approval. The IRB's or IEC's written approval of the protocol and participant informed consent must be obtained and submitted to the Sponsor or designee before commencement of the study (ie, before shipment of the Sponsor-supplied drug or study specific screening activity). The IRB or IEC approval must refer to the study by exact protocol title, number, and version date; identify versions of other documents (eg, informed consent form) reviewed; and state the approval date. The Sponsor will ship drug/notify site once the Sponsor has confirmed the adequacy of site regulatory documentation and, when applicable, the Sponsor has received permission from competent authority to begin the study. Until the site receives drug/notification no protocol activities, including screening, may occur.

Sites must adhere to all requirements stipulated by their respective IRB or IEC. This may include notification to the IRB or IEC regarding protocol amendments, updates to the informed consent form, recruitment materials intended for viewing by participants, local safety reporting requirements, reports and updates regarding the ongoing review of the study at intervals specified by the respective IRB or IEC, and submission of the investigator's final status report to IRB or IEC. All IRB and IEC approvals and relevant documentation for these items must be provided to the Sponsor or its designee.

Participant incentives should not exert undue influence for participation. Payments to participants must be approved by the IRB or IEC and Sponsor.

#### 13.2 Participant Information, Informed Consent, and Participant Authorization

1501J50 Written consent documents will embody the elements of informed consent as described in the Declaration of Helsinki and the ICH Guidelines for GCP and will be in accordance with all applicable laws and regulations. The informed consent form, participant authorization form (if applicable), and participant information sheet (if applicable) describe the planned and permitted uses, transfers, and disclosures of the participant's personal and personal health information for purposes of conducting the study. The informed consent form and the participant information sheet (if applicable) further explain the nature of the study, its objectives, and potential risks and benefits, as well as the date informed consent is given. The informed consent form will detail the requirements of the participant and the fact that he or she is free to withdraw at any time without giving a reason and without prejudice to his or her further medical care.

The investigator is responsible for the preparation, content, and IRB or IEC approval of the informed consent form and, if applicable, the participant authorization form. The informed consent form, participant authorization form (if applicable), and participant information sheet (if applicable) must be approved by both the IRB or IEC and the Sponsor prior to use.

The informed consent form, participant authorization form (if applicable), and participant information sheet (if applicable) must be written in a language fully comprehensible to the prospective participant. It is the responsibility of the investigator to explain the detailed elements of the informed consent form, participant authorization form (if applicable), and participant information sheet (if applicable) to the participant. Information should be given in both oral and written form whenever possible and in the manner deemed appropriate by the IRB or IEC. In the event the participant is not capable of rendering adequate written informed consent, then the participant's legally acceptable representative may provide such consent for the participant in accordance with applicable laws and regulations.

The participant, or the participant's legally acceptable representative, must be given ample opportunity to: (1) inquire about details of the study, and (2) decide whether or not to participate in the study. If the participant, or the participant's legally acceptable representative, determines he or she will participate in the study, then the informed consent form and participant authorization form (if applicable) must be signed and dated by the participant, or the participant's legally acceptable representative, at the time of consent and prior to the participant entering into the study. The participant or the participant's legally acceptable representative should be instructed to sign using their legal names, not nicknames, using blue or black ballpoint ink. The investigator must also sign and date the informed consent form and participant authorization (if applicable) at the time of consent and prior to participant entering into the study; however, the Sponsor may allow a designee of the investigator to sign to the extent permitted by applicable law.

Once signed, the original informed consent form, participant authorization form (if applicable), and participant information sheet (if applicable) will be stored in the investigator's site file. The investigator must document the date the participant signs the informed consent in the participant's medical record. Copies of the signed informed consent form, the signed participant authorization form (if applicable), and participant information sheet (if applicable) shall be given to the participant.

All revised informed consent forms must be reviewed and signed by relevant participants or the relevant participant's legally acceptable representative in the same manner as the original informed consent. The date the revised consent was obtained should be recorded in the participant's medical record, and the participant should receive a copy of the revised informed consent form.

#### 13.3 Participant Confidentiality

The Sponsor and designees affirm and uphold the principle of the participant's right to protection against invasion of privacy. Throughout this study, a participant's source data will only be linked to the Sponsor's clinical study database or documentation via a unique identification number. As permitted by all applicable laws and regulations, limited participant attributes, such as sex, age, or date of birth, and participant initials may be used to verify the participant and accuracy of the participant's unique identification number.

To comply with ICH Guidelines for GCP and to verify compliance with this protocol, the Sponsor requires the investigator to permit its monitor or designee's monitor, representatives from any regulatory authority (eg, FDA, Medicines and Healthcare products Regulatory Agency, Pharmaceuticals and Medical Devices Agency), the Sponsor's designated auditors, and the appropriate IRBs and IECs to review the participant's original medical records (source data or documents), including, but not limited to, laboratory test result reports, ECG reports, admission and discharge summaries for hospital admissions occurring during a participant's study participation, and autopsy reports. Access to a participant's original medical records requires the specific authorization of the participant as part of the informed consent process (see Section 13.2).

Copies of any participant source documents that are provided to the Sponsor must have certain personally identifiable information removed (ie, participant name, address, and other identifier fields not collected on the participant's CRF).

# 13.4 Publication, Disclosure, and Clinical Study Registration Policy

#### 13.4.1 Publication and Disclosure

The investigator is obliged to provide the Sponsor with complete test results and all data derived by the investigator from the study. During and after the study, only the Sponsor may make study information available to other study investigators or to regulatory agencies, except as required by law or regulation. Except as otherwise allowable in the clinical study site agreement, any public disclosure (including publicly accessible websites) related to the protocol or study results, other than study recruitment materials and/or advertisements, is the sole responsibility of the Sponsor.

The Sponsor may publish any data and information from the study (including data and information generated by the investigator) without the consent of the investigator. Manuscript authorship for any peer-reviewed publication will appropriately reflect contributions to the production and review of the document. All publications and presentations must be prepared in accordance with this section and the Clinical Study Site Agreement. In the event of any discrepancy between the protocol and the Clinical Study Site Agreement, the Clinical Study Site Agreement will prevail.

## 13.4.2 Clinical Study Registration

In order to ensure that information on clinical trials reaches the public in a timely manner and to comply with applicable laws, regulations and guidance, Takeda will, at a minimum register all interventional clinical trials it Sponsors anywhere in the world on ClinicalTrials.gov and/or other publicly accessible websites before start of study, as defined in Takeda Policy/Standard. Takeda contact information, along with investigator's city, state (for Americas investigators), country, and recruiting status will be registered and available for public viewing.

For some registries, Takeda will assist callers in locating study sites closest to their homes by providing the investigator name, address, and phone number to the callers requesting trial information. Once participants receive investigator contact information, they may call the site requesting enrollment into the trial. The investigative sites are encouraged to handle the trial inquiries according to their established participant screening process. If the caller asks additional questions beyond the topic of trial enrollment, they should be referred to the Sponsor.

Any investigator who objects to the Sponsor providing this information to callers must provide the Sponsor with a written notice requesting that their information not be listed on the registry site.

## 13.4.3 Clinical Study Results Disclosure

Takeda will post the results of clinical studies on ClinicalTrials.gov or other publicly accessible websites, as required by Takeda Policy/Standard, applicable laws and/or regulations.

# 13.5 Insurance and Compensation for Injury

Each participant in the study must be insured in accordance with the regulations applicable to the site where the participant is participating. If a local underwriter is required, then the Sponsor or Sponsor's designee will obtain clinical study insurance against the risk of injury to study participants. Refer to the study site agreement regarding the Sponsor's policy on participant compensation and treatment for injury. If the investigator has questions regarding this policy, he or she should contact the Sponsor or Sponsor's designee.

#### 14.0 ADMINISTRATIVE AND REFERENCE INFORMATION

#### 14.1 Administrative Information

#### **Study Contact Information** 14.1.1

| Contact Type / Role | Contact |
|---|---|
| Serious adverse event and pregnancy reporting | Pharmacovigilance Takeda Development Center Americas, Inc. E-mail: eupv@tgrd.com Fax: +1-202-315-3560 |
| | licable |
| | "He Vol. |
| | ioject to |
| | and Sur |
| | Se Ouly |
| Mercial | |
| , on Comi | |
| i kor Ac | |
| 14 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
| e <sup>KH</sup> O <sup>X</sup> | |

#### 14.1.2 INVESTIGATOR AGREEMENT

I confirm that I have read and that I understand this protocol, the Investigator's Brochure, package insert and any other product information provided by the Sponsor. I agree to conduct this study in accordance with the requirements of this protocol and also to protect the rights, safety, privacy, and well-being of study participants in accordance with the following:

- The ethical principles that have their origin in the Declaration of Helsinki.
- International Conference on Harmonisation, E6 [R2] Good Clinical Practice: Consolidated Guideline.
- All applicable laws and regulations, including, without limitation, data privacy laws and regulations.
- Regulatory requirements for reporting serious adverse events defined in Section 10.2.9 of this protocol.
- Terms outlined in the study site agreement.
- Responsibilities of the Investigator (Appendix B).

I further authorize that my personal information may be processed and transferred in accordance with the uses contemplated in Appendix D of this protocol.

| Signature of Investigator | Date |
|---------------------------------------------|------|
| Investigator Name (print or type) | |
| Colex | |
| Investigator's Title | |
| Location of Facility (City, State/Provence) | |
| 4080 | |
| Location of Facility (Country) | |
| O, | |

The Sponsor will perform all study-related activities with the exception of those identified in the Study-Related Responsibilities template. The vendors identified for specific study-related activities will perform these activities in full or in partnership with the Sponsor.

14.1.4 List of Abbreviations

AE Adverse event

ALT Alanine aminotransferase

AST Aspartate aminotransferase

AUC Area under the concentration-time curve

AUC<sub>∞</sub> Area under the concentration.

Area under the concentration-time curve from time 0 to infinity  $AUC_{\infty}$ 

 $AUC_{last}$ Area under the concentration-time curve from time 0 to the time of the last quantifiable

concentration

Area under the curve from the last quantifiable concentration to infinity AUC<sub>extrap%</sub>

BID Twice daily **BMI** Body mass index Beats per minute bpm

C-SSRS Columbia-Suicide Severity Rating Scale

Code of Federal Regulations **CFR** CH24H Cholesterol 24S-hydroxylase Confidence interval CI

CL/F Apparent clearance after extravascular administration

Maximum observed concentration  $C_{\text{max}}$ 

Coronavirus disease 2019 COVID-19

Case report form **CRF** Clinical Research Unit **CRU CSR** Clinical study report **CYP** Cytochrome P450 DDI Drug-drug interaction

Developmental and Epileptic Encephalopathies DEE

DS Dravet Syndrome **ECG** Electrocardiogram

**FSH** Follicle stimulating hormone **GCP** Good Clinical Practice **GMR** Geometric mean ratio HBsAg Hepatitis B surface antigen

**HCV** Hepatitis C virus

HIV Human immunodeficiency virus

ΙB Investigator's Brochure **ICF** Informed Consent Form

| ICH | International Council for Harmonisation |
|---|---|
| IEC | Independent Ethics Committee |
| INR | International normalized ratio |
| IRB | Institutional Review Board |
| LFT | Liver function test |
| ln | International normalized ratio Institutional Review Board Liver function test Natural log Lennox Gastaut Syndrome Medical Dictionary for Regulatory Activities® organic-anion-transporting polypeptide P-glycoprotein Physiologically-based PK Pharmacokinetic(s) Pretreatment event Once daily QT interval corrected for heart rate using Fridericia's formula |
| LGS | Lennox Gastaut Syndrome |
| $MedDRA^{\mathbb{R}}$ | Medical Dictionary for Regulatory Activities® |
| OATP | organic-anion-transporting polypeptide |
| P-gp | P-glycoprotein |
| PBPK | Physiologically-based PK |
| PK | Pharmacokinetic(s) |
| PTE | Pretreatment event |
| QD | Once daily |
| QTcF | QT interval corrected for heart rate using Fridericia's formula |
| RNA | Ribonucleic acid Serious adverse event Statistical analysis plan |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SUSAR | Suspected unexpected serious adverse reactions |
| $t_{1/2z}$ | Terminal disposition phase half-life |
| T4 | Immediate release tablets |
| TEAE | Treatment-emergent adverse event |
| $t_{max}$ | Time of first occurrence of C <sub>max</sub> |
| ULN | Upper limit of normal |
| US | United States |
| USA | United States of America |

# 15.0 DATA HANDLING AND RECORD KEEPING

The full details of procedures for data handling will be documented in the Data Management Plan. AEs, medical history, and concurrent conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Drugs will be coded using the World Health Organization Drug Dictionary.

# 15. O CRFs (Electronic and Paper)

Celerion standard CRFs will be supplied. CRFs are produced, stored electronically, and are available to the designated study team members. Each CRF is reviewed and signed by the Investigator. The final signed CRFs are provided to the Sponsor in the format as decided upon between Celerion and the Sponsor (e.g., CD, flashdrive, SFTP). This will be documented in the Data Management Plan (if applicable).

After completion of the entry process, computer logic checks will be run to identify items, such as inconsistent dates, missing data, and questionable values. Queries may be issued by Takeda personnel (or designees) and will be answered by the site.

Corrections are recorded in an audit trail that captures the old information, the new information identification of the person making the correction, the date the correction was made, and the reason for change. Reasons for significant corrections should additionally be included.

The principal investigator must review the CRFs for completeness and accuracy and must sign and date the appropriate CRFs as indicated. Furthermore, the investigator must retain full responsibility for the accuracy and authenticity of all data entered on the CRFs.

After the lock of the clinical study database, any change of, modification of, or addition to the data on the CRFs should be made by the investigator with use of change and modification records of the CRFs. The principal investigator must review the data change for completeness and accuracy, and must sign and date.

CRFs will be reviewed for completeness and acceptability at the study site during periodic visits by study monitors. The Sponsor or its designee will be permitted to review the participant's medical and hospital records pertinent to the study to ensure accuracy of the CRFs. The completed CRFs are the sole property of the Sponsor and should not be made available in any form to third parties, except for authorized representatives of appropriate governmental health or regulatory authorities, without written permission of the Sponsor.

### 15.2 Record Retention

The investigator agrees to keep the records stipulated in Section 15.1 and those documents that include (but are not limited to) the study-specific documents, the identification log of all participating participants, medical records, temporary media such as thermal sensitive paper, source worksheets, all original signed and dated informed consent forms, participant authorization forms regarding the use of personal health information (if separate from the informed consent forms), electronic copy of CRFs, including the audit trail, and detailed records of drug disposition to enable evaluations or audits from regulatory authorities, the Sponsor or its designees. Any source documentation printed on degradable thermal sensitive paper should be photocopied by the site and filed with the original in the participant's chart to ensure long-term legibility. Furthermore, ICH E6 Section 4.9.5 requires the investigator to retain essential documents specified in ICH E6 (Section 8) until at least 2 years after the last approval of a marketing application for a specified drug indication being investigated or, if an application is not approved, until at least 2 years after the investigation is discontinued and regulatory authorities are notified. In addition, ICH E6 Section 4.9.5 states that the study records should be Pretained until an amount of time specified by applicable regulatory requirements or for a time specified in the Clinical Study Site Agreement between the investigator and Sponsor.

Refer to the Clinical Study Site Agreement for the Sponsor's requirements on record retention. The investigator and the head of the institution should contact and receive written approval from the Sponsor before disposing of any such documents.

#### 16.0 REFERENCES

- 1. Kupper, L. L. and Hafner, K.B., How appropriate are popular sample size formulas? Am Stat, 1989. 43(2): 101-105
- 2. TAK-935. Takeda Pharmaceutical Company Ltd. Global Investigator's Brochure. Edition 6, 15 January 2021.
- 3. Rifadin<sup>®</sup> (Rifampin) capsules, Sanofi-Aventis U.S. LLC, full prescribing information (electronic monograph; document revised: 12/2020). Available at https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=036ab68e-5085-4edc-bd83-784b43d64eab.
- 4. Food and Drug Administration: Drug Development and Drug Interactions: Table of Substrates, Inhibitors, and Inducers. Available at: https://www.fda.gov/drugs/developmentapprovalprocess/developmentresources/druginteractionslabeling/ucm093664.htm. (26 September 2016).
- 5. Pang, X., et al., Effects of rifampin and ketoconazole on pharmacokinetics of morinidazole in healthy chinese subjects. Antimicrob Agents Chemother, 2014. **58**(10):5987-93.
- 6. Damayanthi, D., et al., Effects of rifampin, cyclosporine A, and probenecid on the pharmacokinetic profile of canagliflozin, a sodium glucose co-transporter 2 inhibitor, in healthy participants. Int J Clin Pharmacol Ther, 2015. **53**(2):115-28.
- 7. Kasichayanula, S., et al., Effects of rifampin and mefenamic acid on the pharmacokinetics and pharmacodynamics of dapagliflozin. Diabetes Obes Metab, 2013. **15**(3):280-3.
- 8. EMA/425645/2020. European Medicines Regulatory Network approach for the implementation of the CHMP Opinion pursuant to Article 5(3) of Regulation (EC) No 726/2004 for nitrosamine impurities in human medicines; Feb 2021. Available at: https://www.ema.europa.eu/en/documents/referral/nitrosamines-emea-h-a53-1490-assessment-report en.pdf
- 9. Kapetas AJ, Sorich MJ, Rodrigues AD, Rowland A. Guidance for rifampin and midazolam dosing protocols to study intestinal and hepatic cytochrome P450 (CYP) 3A4 induction and de-induction. AAPS J. 2019 Jun 19;21(5):78. doi: 10.1208/s12248-019-0341-y. PMID: 31218462.
- 10. Tran JQ, Kovacs SJ, McIntosh TS, Davis HM, and Martin DE. Morning spot and 24-Hour urinary 6β-hydroxycortisol to cortisol ratios: intraindividual variability and correlation under basal conditions and conditions of CYP 3A4 induction. J Clin Pharmacol. 1999;39:487–94.
- 11. Tortorici MA, Matschke K, Korth-Bradley JM, DiLea C, Lasseter KC. The effect of rifampin on the pharmacokinetics of sirolimus in healthy volunteers. Clin Pharmacol Drug Dev, 2014;3(1):51-56.

#### 17.0 **APPENDICES**

Clinical research studies sponsored by the Sponsor are subject to ICH GCP and all the applicable local laws and regulations. The responsibilities imposed on investigators by the FDA are summarized in the "Statement of Investigator" (Fermi Signed hoff). signed before the investigator may participate in this study.

The investigator agrees to assume the following responsibilities by signing a Form FDA 1572:

- 1. Conduct the study in accordance with the protocol.
- 2. Personally conduct or supervise the staff that will assist in the protocol.
- 3. If the investigator/institution retains the services of any individual or party to perform trialrelated duties and functions, the investigator/institution should ensure that this individual or party is qualified to perform those trial-related duties and functions and should implement procedures to ensure the integrity of the trial-related duties and functions performed and any data generated.
- 4. Ensure that study related procedures, including study specific (nonroutine/nonstandard panel) screening assessments are NOT performed on potential participants, prior to the receipt of written approval from relevant governing bodies/authorities.
- 5. Ensure that all colleagues and employees assisting in the conduct of the study are informed of these obligations.
- 6. Secure prior approval of the study and any changes by an appropriate IRB/IEC that conform to 21 CFR Part 56, ICH, and local regulatory requirements.
- 7. Ensure that the IRB/IEC will be responsible for initial review, continuing review, and approval of the protocol. Promptly report to the IRB/IEC all changes in research activity and all anticipated risks to participants. Make at least yearly reports on the progress of the study to the IRB/IEC, and issue a final report within 3 months of study completion.
- 8. Ensure that requirements for informed consent, as outlined in 21 CFR Part 50, ICH and local regulations, are met.
- 9. Obtain valid informed consent from each participant who participates in the study, and document the date of consent in the participant's medical chart. Valid informed consent is the most current version approved by the IRB/IEC. Each informed consent form should contain a participant authorization section that describes the uses and disclosures of a participant's personal information (including personal health information) that will take place in connection with the study. If an informed consent form does not include such a participant authorization, then the investigator must obtain a separate participant authorization form from each participant or the participant's legally acceptable representative.
- 10. Prepare and maintain adequate case histories of all persons entered into the study, including CRFs, hospital records, laboratory results, etc, and maintain these data for a minimum of

- 2 years following notification by the Sponsor that all investigations have been discontinued or that the regulatory authority has approved the marketing application. The investigator should contact and receive written approval from the Sponsor before disposing of any such documents.
- 11. Allow possible inspection and copying by the regulatory authority of GCP-specified essential documents.
- 12. Maintain current records of the receipt, administration, and disposition of Sponsor-supplied drugs, and return all unused Sponsor-supplied drugs to the Sponsor.
- of an SA, of an SA, of an SA, the state of t 13. Report adverse reactions to the Sponsor promptly. In the event of an SAE notify the Sponsor

provided to each participant:

... the purposes of the research.

... the expected duration of the participant's participation.

4. A description of the procedures to be followed, including invasive procedures.

5. The identification of any procedures that are experimental.

6. The estimated number of participants involved in the study.

7. A description of the participant's response.

- 9. A statement describing the treatment(s) and the probability for random assignment to each treatment.
- 10. A description of the possible side effects of the treatment that the participant may receive.
- 11. A description of any reasonably foreseeable risks or discomforts to the participant and, when applicable, to an embryo, fetus, or nursing infant.
- 12. A description of any benefits to the participant or to others that reasonably may be expected from the research. When there is no intended clinical benefit to the participant, the participant should be made aware of this.
- 13. Disclosures of appropriate alternative procedures or courses of treatment, if any, that might be advantageous to the participant and their important potential risks and benefits.
- 14. A statement describing the extent to which confidentiality of records identifying the participant will be maintained, and a note of the possibility that regulatory agencies, auditor(s), IRB/IEC, and the monitor may inspect the records. By signing a written informed consent form, the participant or the participant's legally acceptable representative is authorizing such access.
- 15. For research involving more than minimal risk, an explanation as to whether any compensation and an explanation as to whether any medical treatments are available if injury occurs and, if so, what they consist of or where further information may be obtained.
- 16. The anticipated prorated payment(s), if any, to the participant for participating in the study.
- 7. The anticipated expenses, if any, to the participant for participating in the study.
- 18. An explanation of whom to contact for answers to pertinent questions about the research (investigator), participant's rights, and IRB/IEC and whom to contact in the event of a research-related injury to the participant.

- 19. A statement that participation is voluntary, that refusal to participate will involve no penalty or loss of benefits to which the participant otherwise is entitled, and that the participant or the participant's legally acceptable representative may discontinue participation at any time without penalty or loss of benefits to which the participant is otherwise entitled.
- 20. The consequences of a participant's decision to withdraw from the research and procedures for orderly termination of participation by the participant.
- 21. A statement that the participant or the participant's legally acceptable representative will be informed in a timely manner if information becomes available that may be relevant to the participant's willingness to continue participation in the study.
- 22. The foreseeable circumstances or reasons under which the participant's participation in the study may be terminated.
- 23. A written participant authorization (either contained within the informed consent form or provided as a separate document) describing to the participant the contemplated and permissible uses and disclosures of the participant's personal information (including personal health information) for purposes of conducting the study. The participant authorization must contain the following statements regarding the uses and disclosures of the participant's personal information:
  - a) that personal information (including personal health information) may be processed by or transferred to other parties in other countries for clinical research and safety reporting purposes, including, without limitation, to the following: (1) Takeda, its affiliates, and licensing partners; (2) business partners assisting Takeda, its affiliates, and licensing partners; (3) regulatory agencies and other health authorities; and (4) IRBs/IECs;
  - b) it is possible that personal information (including personal health information) may be processed and transferred to countries that do not have data protection laws that offer participants the same level of protection as the data protection laws within this country; however, Takeda will make every effort to keep your personal information confidential, and your name will not be disclosed outside the clinic unless required by law;
  - c) that personal information (including personal health information) may be added to Takeda's research databases for purposes of developing a better understanding of the safety and effectiveness of the study medication(s), studying other therapies for patients, developing a better understanding of disease, and improving the efficiency of future clinical studies;
  - that participants agree not to restrict the use and disclosure of their personal information (including personal health information) upon withdrawal from the study to the extent that the restricted use or disclosure of such information may impact the scientific integrity of the research; and
  - e) that the participant's identity will remain confidential in the event that study results are published.
- 24. Regular pregnancy tests will be performed throughout the study for all female participants.

- end in a sed

## **Appendix C** Investigator Consent to the Use of Personal Information

Takeda will collect and retain personal information of investigator, including his or her name, address, and other personally identifiable information. In addition, investigator's personal information may be transferred to other parties located in countries throughout the world (eg. the United Kingdom, United States, and Japan), including the following:

- Takeda, its affiliates, and licensing partners.
- Business partners assisting Takeda, its affiliates, and licensing partners.
- Regulatory agencies and other health authorities.
- IRBs and IECs.

Investigator's personal information may be retained, processed, and transferred by Takeda and these other parties for research purposes including the following:

- Assessment of the suitability of investigator for the study and/or other clinical studies.
- Management, monitoring, inspection, and audit of the study.
- Analysis, review, and verification of the study results.
- Safety reporting and pharmacovigilance relating to the study.
- Preparation and submission of regulatory filings, correspondence, and communications to regulatory agencies relating to the study.
- Preparation and submission of regulatory filings, correspondence, and communications to regulatory agencies relating to other medications used in other clinical studies that may contain the same chemical compound present in the study medication.
- Inspections and investigations by regulatory authorities relating to the study.
- Self-inspection and internal audit within Takeda, its affiliates, and licensing partners.
- Archiving and audit of study records.
- Posting investigator site contact information, study details and results on publicly accessible clinical trial registries, databases, and websites.

Investigator's personal information may be transferred to other countries that do not have data protection laws that offer the same level of protection as data protection laws in investigator's own country.

Investigator acknowledges and consents to the use of his or her personal information by Takeda and other parties for the purposes described above.

# Appendix D Pregnancy and Contraception **Contraception and Pregnancy Avoidance Procedure**

Male Participants

Soluse From signing of informed consent, throughout the duration of the study, and for 90 days after last dose of study drug, nonsterilized\* male participants who are sexually active with a female partner of childbearing potential\*\* must use barrier contraception (eg. condom with or without spermicidal cream or jelly). In addition, they must be advised not to donate sperm during this period. Total abstinence (no sexual intercourse) may be considered an acceptable method of birth control if it agrees with his preferred and usual lifestyle.

Female Participants and Their Male Partners

Only women of non-childbearing potential will be included in this study. A female of non-childbearing potential, must have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

- hysteroscopic sterilization;
- bilateral tubal ligation or bilateral salpingectomy;
- hysterectomy;
- bilateral oophorectomy;

or be postmenopausal with amenorrhea for at least 1 year prior to the first dosing and FSH serum levels consistent with postmenopausal status\*\*.

Definitions and Procedures for Contraception and Pregnancy Avoidance

The following definitions apply for contraception and pregnancy avoidance procedures.

- \* Sterilized males should be at least 1 year post-bilateral vasectomy and have confirmed that they have obtained documentation of the absence of sperm in the ejaculate or have had bilateral orchidectomy.
- \*\*A woman is considered a woman of childbearing potential (WOCBP), ie, fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range (FSH >40 IU/L) may be used to confirm a post-menopausal state in younger women (eg, those <45 year old) or women who are not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

General Guidance With Respect to the Avoidance of Pregnancy

Such guidance should include a reminder of the following:

contraceptive requirements of the study.

- reasons for use of barrier methods (ie, condom) in males with pregnant partners.
- assessment of participant compliance through questions such as:
  - Have you used the contraception consistently and correctly since the last visit?
  - Have you forgotten to use contraception since the last visit?

#### **Pregnancy**

Women of childbearing potential will not be included in this study.

cable reims of Use If any participant is found to be pregnant during the study she should be withdrawn and any sponsor-supplied drug should be immediately discontinued. In addition, any pregnancies in the partner of a male participant during the study or for 90 days after the last dose, should also be recorded following authorization from the participant's partner.

If the female participant and/or female partner of a male participant agrees to the primary care physician being informed, the investigator should notify the primary care physician that the female participant and/or female partner of the participant was participating in a clinical study at the time she became pregnant and provide details of the study drug the participant received (blinded or unblinded, as applicable).

All pregnancies, including female partners of male participants, in participants on active study drug (including comparator, if applicable) will be followed up to final outcome, using the Property of Takeda. For Won-Commercial pregnancy form. Pregnancies will remain blinded to the study team. The outcome, including any premature termination, must be reported to the sponsor. An evaluation after the birth of the child

# ELECTRONIC SIGNATURES

| | Signed by | Meaning of Signature | Server Date (dd-MMM-yyyy HH:mm 'UTC') |
|---|---|---|---|
| | | Biostatistics Approval | (dd-MMM-yyyy HH:mm 'UTC')<br>23-Aug-2021 15:00 UTC |
| | | Clinical Approval | 23-Aug-2021 15:50 UTC |
| | | Clinical Pharmacology Approval | 23-Aug-2021 20:25 UTC |
| Prope | Signed by Signed by Signed by | percial Use Only and Subject. | |